CLINICAL TRIAL: NCT03135834
Title: A PHASE 3, RANDOMIZED, ACTIVE-CONTROLLED, OBSERVER-BLINDED STUDY TO ASSESS THE IMMUNOGENICITY, SAFETY, AND TOLERABILITY OF BIVALENT RLP2086 WHEN ADMINISTERED AS A 2-DOSE REGIMEN AND A FIRST-IN-HUMAN STUDY TO DESCRIBE THE IMMUNOGENICITY, SAFETY, AND TOLERABILITY OF A BIVALENT RLP2086-CONTAINING PENTAVALENT VACCINE (MENABCWY) IN HEALTHY SUBJECTS>=10 TO <26 YEARS OF AGE
Brief Title: A Trial to Describe the Immunogenicity and Safety of 2 Doses of Bivalent rLP2086 (Trumenba) and a Pentavalent Meningococcal Vaccine in Healthy Subjects >=10 to <26 Years of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1971057; 2016-004421-17 (EudraCT Number)
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Meningococcal Vaccine
MeSH Terms: interventions — Sodium Chloride; factor H-binding protein, Neisseria meningitidis; MenACWY-CRM vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (ACWY Naive subjects, MenABCWY/Saline) (Experimental): ACWY Naive subjects, MenABCWY/Saline
  Interventions: Biological: MenABCWY; Biological: Saline
- Group 2 (ACWY Naive subjects, rLP2086/MenACWY-CRM) (Experimental): ACWY Naive subjects, rLP2086/MenACWY-CRM
  Interventions: Biological: rLP2086; Biological: MenACWY-CRM
- Group 3 (ACWY Experienced subjects, MenABCWY/Saline) (Experimental): ACWY Experienced subjects, MenABCWY/Saline
  Interventions: Biological: MenABCWY; Biological: Saline
- Group 4 (ACWY Experienced subjects, rLP2086/MenACWY-CRM) (Experimental): ACWY Experienced subjects, rLP2086/MenACWY-CRM
  Interventions: Biological: rLP2086; Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenABCWY — N meningitidis group A, B, C, W, and Y vaccine
  Arms: Group 1 (ACWY Naive subjects, MenABCWY/Saline); Group 3 (ACWY Experienced subjects, MenABCWY/Saline)
Biological: Saline — Placebo
  Arms: Group 1 (ACWY Naive subjects, MenABCWY/Saline); Group 3 (ACWY Experienced subjects, MenABCWY/Saline)
Biological: rLP2086 — Bivalent recombinant lipoprotein 2086 vaccine
  Arms: Group 2 (ACWY Naive subjects, rLP2086/MenACWY-CRM); Group 4 (ACWY Experienced subjects, rLP2086/MenACWY-CRM)
Biological: MenACWY-CRM — meningococcal group A, C, W-135, and Y conjugate vaccine
  Arms: Group 2 (ACWY Naive subjects, rLP2086/MenACWY-CRM); Group 4 (ACWY Experienced subjects, rLP2086/MenACWY-CRM)

SUMMARY:
This study is examining safety and immunogenicity of 2 doses of Trumenba administered on a 0-,6- month schedule. This trial is also studying safety and immunogenicity of a meningococcal pentavalent vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged >=10 and <26 years at the time of enrollment.
* Healthy subject as determined by medical history, physical examination, and judgment of the investigator.
* Negative urine pregnancy test for all female subjects.
* Subjects who have not received, or who have received no more than 1 prior dose within the past 4 years, of a vaccine containing 1 or more ACWY serogroup

Exclusion Criteria:

* Previous vaccination with any meningococcal serogroup B or purely polysaccharide (nonconjugate) meningococcal vaccine.
* Subjects receiving any allergen immunotherapy with a nonlicensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
* A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired defects in B cell function, those receiving chronic systemic (oral, intravenous, or intramuscular) corticosteroid therapy, or those receiving immunosuppressive therapy. Subjects in the United States with terminal complement deficiency are excluded from participation in this study.
* Significant neurological disorder or history of seizure (excluding simple febrile seizure).
* Current chronic use of systemic antibiotics.
* Received any investigational vaccines, drugs, or devices within 28 days before administration of the first study vaccination.
* Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1610 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- United States (57):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Optimal Research, LLC, Huntsville, Alabama
  - Synexus Clinical Research US, Inc./Fountain Hills Family Practice, P.C., Fountain Hills, Arizona
  - Clinical Research Consortium, Tempe, Arizona
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - Paradigm Clinical Research Centers, Inc., La Mesa, California
  - California Research Foundation, San Diego, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Optimal Research, LLC, Melbourne, Florida
  - Meridian Clinical Research LLC, Savannah, Georgia
  - Optimal Research, Peoria, Illinois
  - Meridian Clinical Research, Sioux City, Iowa
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Alliance For Multispecialty Research (AMR), Wichita, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Horizon Research Group of Opelousas, LLC, Eunice, Louisiana
  - ACC Pediatric Research, Haughton, Louisiana
  - Methodist Physicians Clinic/CCT Research, Fremont, Nebraska
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Binghamton, New York
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc, Endwell, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Meridian Clinical Research, LLC, Vestal, New York
  - Regional Clinical Research, Inc, Vestal, New York
  - Capitol Pediatrics & Adolescent Center PLLC, Raleigh, North Carolina
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Velocity Clinical Research, Inc., Cleveland, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - Ohio Pediatric Research Association, Inc., Dayton, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Liberty Family Practice, Erie, Pennsylvania
  - Charleston Pediatrics, PA, Charleston, South Carolina
  - PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Texas Health Care, PLLC, Fort Worth, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Benchmark Research, Fort Worth, Texas
  - Acrc Trials, Plano, Texas
  - North Texas Family Medicine, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - J. Lewis Research Inc. / Foothill Family Clinic Draper, Draper, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
- Czechia (2):
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - MEDICENTRUM 6 s.r.o. - Ordinace praktickeho lekare pro deti a dorost, Prague
- Finland (10):
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Jarvenpaa Vaccine Research Clinic, Jarvenpaa
  - Kokkola Vaccine Research Clinic, Kokkola
  - Oulu Vaccine Research Clinic, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Seinajoki Vaccine Research Clinic, Seinäjoki
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Clinic, Turku
- Poland (3):
  - Jerzy Brzostek Prywatny Gabinet Lekarski, Dębica
  - Hanna Czajka Indywidualna Specjalistyczna Praktyka Lekarska, Krakow
  - Oddzial Pediatrii i Neurologii Dzieciecej, Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Peterson J, Drazan D, Moughan B, Maguire JD, Zolotas L, Maansson R, O'Neill R, Peyrani P, Jodar L, Gruber WC, Anderson AS, Beeslaar J. Randomized trial showing persistence of hSBA titers elicited by a pentavalent meningococcal MenABCWY vaccine for up to 4 years following a primary series and safety and immunogenicity of a booster dose. Vaccine. 2025 Jan 1;43(Pt 1):126469. doi: 10.1016/j.vaccine.2024.126469. Epub 2024 Nov 8. PMID 39520893
- [Derived] Peterson J, Drazan D, Czajka H, Maguire J, Pregaldien JL, Seppa I, Maansson R, O'Neill R, Balmer P, Jodar L, Jansen KU, Anderson AS, Perez JL, Beeslaar J. Immunogenicity and safety of a pentavalent meningococcal ABCWY vaccine in adolescents and young adults: an observer-blind, active-controlled, randomised trial. Lancet Infect Dis. 2023 Dec;23(12):1370-1382. doi: 10.1016/S1473-3099(23)00191-3. Epub 2023 Aug 11. PMID 37579773
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1971057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had 2 stages: 1 and 2. Study was conducted at 68 sites in Stage 1, with 39 of those sites participating in Stage 2. Participants were randomized as ACWY-naive and ACWY-experienced (received 1 prior dose of a vaccine containing 1 or more ACWY groups greater than or equal to [>=] 4 years prior to randomization).
Pre-assignment Details: A total of 1610 participants were randomized in this study, out of which 10 withdrew before vaccination.
Groups:
- Group 1: MenABCWY + Saline (ACWY-Naive): Stage 1: ACWY-naive participants were randomized to receive an intramuscular injection of 0.5 milliliter (mL) of Neisseria meningitidis groups A, B, C, W, and Y vaccine (MenABCWY) and 0.5 mL of saline at Month 0, participants received 0.5 mL of MenABCWY vaccine intramuscularly at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants had blood drawn for antibody persistence at Month 18, 30, 42. There was a blood draw at Month 0, Month 6 and Month 54 before Vaccination 1, 2 and Booster vaccination. Post vaccination blood draw happened at 1 month after Vaccination 1, 2 and Booster vaccination. Participants received 0.5 mL of MenABCWY vaccine (booster vaccination) intramuscularly at Month 54. There was a safety follow-up 6 months after Vaccination 2 in Stage 1 (Visit 5) and 6 months after Booster Vaccination in Stage 2 (Visit 12).
- Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive): Stage 1: ACWY-naive participants were randomized to receive an intramuscular injection of 0.5 mL bivalent recombinant lipoprotein 2086 (rLP2086) vaccine and 0.5 mL of meningococcal group A, C, W-135, and Y conjugate vaccine (MenACWY-CRM) at Month 0. Participants received 0.5 mL of bivalent rLP2086 vaccine at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants had blood drawn for antibody persistence at Month 18, 30, 42. There was a blood draw at Month 0, Month 6 and Month 54 before Vaccination 1, 2 and Booster vaccination. Post vaccination blood draw happened at 1 month after Vaccination 1, 2 and Booster vaccination. Participants received intramuscularly injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL of MenACWY-CRM vaccine (booster vaccination) at Month 54. There was a safety follow-up 6 months after Vaccination 2 in Stage 1 (Visit 5) and 6 months after Booster Vaccination in Stage 2 (Visit 12).
- Group 3: MenABCWY + Saline (ACWY-Experienced): Stage 1: ACWY-experienced participants were randomized to receive an intramuscular injection of 0.5 milliliter (mL) of Neisseria meningitidis groups A, B, C, W, and Y vaccine (MenABCWY) and 0.5 mL of saline at Month 0, participants received 0.5 mL of MenABCWY vaccine intramuscularly at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants had blood drawn for antibody persistence at Month 18, 30, 42. There was a blood draw at Month 0, Month 6 and Month 54 before Vaccination 1, 2 and Booster vaccination. Post vaccination blood draw happened at 1 month after Vaccination 1, 2 and Booster vaccination. Participants received 0.5 mL of MenABCWY vaccine (booster vaccination) intramuscularly at Month 54. There was a safety follow-up 6 months after Vaccination 2 in Stage 1 (Visit 5) and 6 months after Booster Vaccination in Stage 2 (Visit 12).
- Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced): Stage 1: ACWY-experienced participants were randomized to receive an intramuscular injection of 0.5 mL bivalent recombinant lipoprotein 2086 (rLP2086) vaccine and 0.5 mL of meningococcal group A, C, W-135, and Y conjugate vaccine (MenACWY-CRM) at Month 0. Participants received 0.5 mL of bivalent rLP2086 vaccine at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants had blood drawn for antibody persistence at Month 18, 30, 42. There was a blood draw at Month 0, Month 6 and Month 54 before Vaccination 1, 2 and Booster vaccination. Post vaccination blood draw happened at 1 month after Vaccination 1, 2 and Booster vaccination. Participants received intramuscularly injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL of MenACWY-CRM vaccine (booster vaccination) at Month 54. There was a safety follow-up 6 months after Vaccination 2 in Stage 1 (Visit 5) and 6 months after Booster Vaccination in Stage 2 (Visit 12).
Period: Stage 1
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Started | 272 | 537 | 272 | 529
Vaccination 1 at Month 0 | 272 | 534 | 271 | 523
Vaccination 2 at Month 6 | 242 | 469 | 244 | 477
Completed | 233 (Completed Vaccination) | 462 (Completed Vaccination) | 232 (Completed Vaccination) | 463 (Completed Vaccination)
Not Completed | 39 | 75 | 40 | 66
Not completed — Adverse Event | 1 | 2 | 2 | 1
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 17 | 24 | 21 | 38
Not completed — No longer met eligibility criteria | 1 | 6 | 2 | 5
Not completed — Other | 0 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 4 | 2 | 4
Not completed — Protocol Violation | 1 | 1 | 2 | 1
Not completed — Withdrawal by parent/guardian | 2 | 10 | 2 | 1
Not completed — Withdrawal by Subject | 16 | 22 | 7 | 10
Not completed — Randomized but not Vaccinated | 0 | 3 | 1 | 6
Period: Stage 2
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Started | 114 (Eligible participants entered Stage 2.) | 65 (Eligible participants entered Stage 2.) | 101 (Eligible participants entered Stage 2.) | 73 (Eligible participants entered Stage 2.)
Antibody Persistence: Blood Draw Month18 | 114 | 63 | 53 | 23
Antibody Persistence: Blood Draw Month 30 | 104 | 61 | 96 | 71
Antibody Persistence: Blood Draw Month 42 | 97 | 55 | 97 | 68
Received Booster Vaccination | 67 | 40 | 77 | 58 (Two participants were not included in summary of demographics (safety population) for stage 2 since they were of mixed regimen (received MenABCWY at the booster vaccination instead of bivalent rLP2086 + MenACWY-CRM as randomized).)
Completed (Completed Stage 2) | 67 (Completed Stage 2) | 38 (Completed Stage 2) | 77 (Completed Stage 2) | 58 (Completed Stage 2)
Not Completed | 47 | 27 | 24 | 15
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Withdrawn Before Booster Vaccination | 46 | 24 | 24 | 15
Not completed — Did not receive Booster Vaccination | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population for Stage 1 included participants who had received at least 1 dose of investigational product during Stage 1 and for whom safety data were available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced) | Total
Number analyzed (Participants) | 272 | 534 | 271 | 523 | 1600
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Stage 1 safety population and Booster safety population were evaluated for baseline characteristics for Stage 1 and Stage 2, respectively. 'Number Analyzed' signifies number of participants evaluable for the respective stages. Two participants were not included in summary of demographics (safety population) for stage 2 since they were of mixed regimen (received MenABCWY at the booster vaccination instead of bivalent rLP2086 + MenACWY-CRM as randomized).
  Years
    Stage 1 | 16.0 (5.67) | 16.5 (5.81) | 17.7 (3.57) | 17.8 (3.66) | 17.1 (4.87)
    Stage 2: number analyzed (Participants) | 67 | 40 | 77 | 56 | 240
    Stage 2 | 19.1 (5.36) | 18.5 (5.51) | 20.8 (3.73) | 21.1 (4.11) | 20.4 (4.72)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Stage 1 safety population and Booster safety population were evaluated for baseline characteristics for Stage 1 and Stage 2, respectively. 'Number Analyzed' signifies number of participants evaluable for the respective stages. Two participants were not included in summary of demographics (safety population) for stage 2 since they were of mixed regimen (received MenABCWY at the booster vaccination instead of bivalent rLP2086 + MenACWY-CRM as randomized).
  Participants
    Stage 1: Female | 144 | 333 | 152 | 289 | 918
    Stage 1: Male | 128 | 201 | 119 | 234 | 682
    Stage 2: number analyzed (Participants) | 67 | 40 | 77 | 56 | 240
    Stage 2: Female | 28 | 26 | 47 | 29 | 130
    Stage 2: Male | 39 | 14 | 30 | 27 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Stage 1 safety population and Booster safety population were evaluated for baseline characteristics for Stage 1 and Stage 2, respectively. 'Number Analyzed' signifies number of participants evaluable for the respective stages. Two participants were not included in summary of demographics (safety population) for stage 2 since they were of mixed regimen (received MenABCWY at the booster vaccination instead of bivalent rLP2086 + MenACWY-CRM as randomized).
  Participants
    Stage 1: Hispanic or Latino | 35 | 73 | 24 | 61 | 193
    Stage 1: Not Hispanic or Latino | 236 | 461 | 246 | 461 | 1404
    Stage 1: Unknown or Not Reported | 1 | 0 | 1 | 1 | 3
    Stage 2: number analyzed (Participants) | 67 | 40 | 77 | 56 | 240
    Stage 2: Hispanic or Latino | 6 | 3 | 3 | 1 | 13
    Stage 2: Not Hispanic or Latino | 61 | 37 | 74 | 55 | 227
    Stage 2: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Stage 1 safety population and Booster safety population were evaluated for baseline characteristics for Stage 1 and Stage 2, respectively. 'Number Analyzed' signifies number of participants evaluable for the respective stages. Two participants were not included in summary of demographics (safety population) for stage 2 since they were of mixed regimen (received MenABCWY at the booster vaccination instead of bivalent rLP2086 + MenACWY-CRM as randomized).
  Participants
    Stage 1: American Indian or Alaska Native | 10 | 13 | 6 | 20 | 49
    Stage 1: Asian | 1 | 4 | 3 | 8 | 16
    Stage 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Stage 1: Black or African American | 27 | 53 | 25 | 60 | 165
    Stage 1: White | 234 | 464 | 237 | 435 | 1370
    Stage 1: More than one race | 0 | 0 | 0 | 0 | 0
    Stage 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
    Stage 2: number analyzed (Participants) | 67 | 40 | 77 | 56 | 240
    Stage 2: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Stage 2: Asian | 0 | 0 | 0 | 1 | 1
    Stage 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Stage 2: Black or African American | 5 | 3 | 4 | 2 | 14
    Stage 2: White | 59 | 37 | 72 | 53 | 221
    Stage 2: More than one race | 0 | 0 | 0 | 0 | 0
    Stage 2: Unknown or Not Reported | 3 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Stage1: Percentage of Participants Achieving Serum Bactericidal Assay Using Human Complement (hSBA) Titer Level >= Lower Limit of Quantitation (LLOQ) for All 4 Primary Test Strains Combined 1 Month After Vaccination 2 (Group 2 and 4 Combined)
Description: Percentage of participants who achieved an hSBA titer >= LLOQ for all 4 primary MenB test strains combined (LLOQ was 1:16 for A22 and 1:8 for A56, B24, and B44) was reported in this outcome. Analysis for this outcome measure was planned for combined Group 2 and 4.
Time Frame: 1 month after Vaccination 2
Population: Stage 1 evaluable immunogenicity population(EIP)=all participants randomized to study group of interest,received all investigational products as randomized,had blood drawn for assay testing in required time frames at Months 0 and 7,had valid and determinate assay results,received no prohibited vaccines/treatment,had no major protocol violation determined by medical monitor.'Number of Participants Analyzed'=participants with valid and determinate hSBA results on all 4 strains at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM): Stage 1: ACWY-naive and experienced participants received an intramuscular injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL MenACWY-CRM vaccine at Month 0. Participants received 0.5 mL of bivalent rLP2086 vaccine at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received an intramuscular injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL MenACWY-CRM vaccine at Month 54.
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 814
Percentage of participants | 74.3 [71.2 to 77.3]

2. Primary Outcome: Stage1: Percentage of Participants With Fold Rise >=4 in hSBA for Each of the 4 Primary MenB Test Strains From Baseline to 1 Month After Vaccination 2 (Group 2 and 4 Combined)
Description: The 4-fold increase: a) participants with baseline hSBA titer below limit of detection (LOD or an hSBA titer <1:4), response was defined as hSBA titer >=1:16 or LLOQ (whichever titer is higher); b) Participants with baseline hSBA titer >= LOD and < LLOQ, response was defined as hSBA titer >= 4 times the LLOQ; c) participants with baseline hSBA titer >= LLOQ, response was defined as hSBA titer >=4 times baseline titer. Four primary MenB test strains were PMB80 (A22), PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44). Analysis for this outcome measure was planned for combined Group 2 and 4.
Time Frame: From Baseline (blood draw prior to Vaccination 1) to 1 month after Vaccination 2
Population: Stage 1 EIP analyzed. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. "Number Analyzed": participants with valid and determinate hSBA titers for given strain at both specified time point and baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 864
Percentage of participants
  PMB80 (A22): number analyzed (Participants) | 827
  PMB80 (A22) | 73.8 [70.6 to 76.7]
  PMB2001 (A56): number analyzed (Participants) | 823
  PMB2001 (A56) | 95.0 [93.3 to 96.4]
  PMB2948 (B24): number analyzed (Participants) | 835
  PMB2948 (B24) | 67.4 [64.1 to 70.6]
  PMB2707 (B44): number analyzed (Participants) | 850
  PMB2707 (B44) | 86.4 [83.9 to 88.6]

3. Primary Outcome: Stage1: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1 (Group 2 and 4 Combined)
Description: Local reactions (redness, swelling, and pain) at the site of investigational product administration were recorded in e-diary. Redness and swelling were measured and recorded in caliper units. Each caliper unit represented 0.5 cm. Redness and swelling were graded as mild (>2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm) and severe (>10.0 cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity).
Time Frame: 7 days after Vaccination 1
Population: Vaccination 1 safety population included participants who received the first dose of investigational product (MenABCWY+saline or bivalent rLP2086+MenACWY-CRM) at Visit 1 (Month 0), and for whom safety information from Visit 1 (Month 0) to prior to Visit 3 (Month 6) was available. Here, 'Overall Number of participants Analyzed' signifies number of participants with known values. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1044
Percentage of participants
  Redness: Any | 16.9 [14.6 to 19.3]
  Redness: Mild | 6.8 [5.3 to 8.5]
  Redness: Moderate | 8.0 [6.5 to 9.9]
  Redness: Severe | 2.0 [1.2 to 3.1]
  Swelling: Any | 17.0 [14.7 to 19.4]
  Swelling: Mild | 9.8 [8.0 to 11.7]
  Swelling: Moderate | 6.9 [5.4 to 8.6]
  Swelling: Severe | 0.3 [0.1 to 0.8]
  Pain at injection site: Any | 85.0 [82.6 to 87.1]
  Pain at injection site: Mild | 41.2 [38.2 to 44.2]
  Pain at injection site: Moderate | 39.1 [36.1 to 42.1]
  Pain at injection site: Severe | 4.7 [3.5 to 6.2]

4. Primary Outcome: Stage1: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2 (Group 2 and 4 Combined)
Description: as for outcome 3
Time Frame: 7 days after Vaccination 2
Population: Vaccination 2 safety population included participants who received the second dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 3 (Month 6), and for whom safety information from Visit 3 (Month 6) up to and including Visit 4 (month 7) was available. Here, 'Overall Number of Participants Analyzed' signifies number of participants with known values. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 903
Percentage of participants
  Redness: Any | 14.7 [12.5 to 17.2]
  Redness: Mild | 5.2 [3.8 to 6.9]
  Redness: Moderate | 8.4 [6.7 to 10.4]
  Redness: Severe | 1.1 [0.5 to 2.0]
  Swelling: Any | 14.3 [12.1 to 16.7]
  Swelling: Mild | 6.4 [4.9 to 8.2]
  Swelling: Moderate | 7.5 [5.9 to 9.4]
  Swelling: Severe | 0.3 [0.1 to 1.0]
  Pain at injection site: Any | 82.2 [79.5 to 84.6]
  Pain at injection site: Mild | 38.9 [35.7 to 42.1]
  Pain at injection site: Moderate | 37.9 [34.7 to 41.1]
  Pain at injection site: Severe | 5.4 [4.0 to 7.1]

5. Primary Outcome: Stage1: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1 (Group 2 and 4 Combined)
Description: Systemic events fever, vomiting, diarrhea, headache, fatigue, chills, muscle pain other than muscle pain at the injection site, and joint pain were recorded by using an e-diary. Fever was defined as >=38.0 degree Celsius (C) and categorized to 38.0 to 38.4 degree C, 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and >40.0 degree C. Headache, fatigue, chills, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily activity). Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required IV hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 in 24 hours).
Time Frame: 7 days after Vaccination 1
Population: Vaccination 1 safety population included participants who received the first dose of investigational product (MenABCWY+saline or bivalent rLP2086+MenACWY-CRM) at Visit 1 (Month 0), and for whom safety information from Visit 1 (Month 0) to prior to Visit 3 (Month 6) was available. Here, "Overall Number of Participants Analyzed": number of participants with known values. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1044
Percentage of participants
  Fever: >= 38.0 degree C | 6.7 [5.3 to 8.4]
  Fever: 38.0 to 38.4 degree C | 4.0 [2.9 to 5.4]
  Fever: 38.5 to 38.9 degree C | 2.1 [1.3 to 3.2]
  Fever: 39.0 to 40.0 degree C | 0.6 [0.2 to 1.2]
  Fever: > 40.0 degree C | 0.0 [0.0 to 0.4]
  Fatigue: Any | 51.9 [48.8 to 55.0]
  Fatigue: Mild | 25.4 [22.8 to 28.1]
  Fatigue: Moderate | 23.7 [21.1 to 26.4]
  Fatigue: Severe | 2.9 [1.9 to 4.1]
  Headache: Any | 46.5 [43.4 to 49.5]
  Headache: Mild | 25.1 [22.5 to 27.8]
  Headache: Moderate | 19.0 [16.6 to 21.5]
  Headache: Severe | 2.4 [1.6 to 3.5]
  Chills: Any | 18.5 [16.2 to 21.0]
  Chills: Mild | 11.5 [9.6 to 13.6]
  Chills: Moderate | 5.7 [4.4 to 7.3]
  Chills: Severe | 1.2 [0.7 to 2.1]
  Vomiting: Any | 3.7 [2.7 to 5.1]
  Vomiting: Mild | 2.9 [1.9 to 4.1]
  Vomiting: Moderate | 0.9 [0.4 to 1.6]
  Vomiting: severe | 0.0 [0.0 to 0.4]
  Diarrhea: Any | 14.1 [12.0 to 16.3]
  Diarrhea: Mild | 10.7 [8.9 to 12.8]
  Diarrhea: Moderate | 3.3 [2.3 to 4.5]
  Diarrhea: Severe | 0.1 [0.0 to 0.5]
  Muscle pain: Any | 28.4 [25.7 to 31.3]
  Muscle pain: Mild | 15.8 [13.6 to 18.2]
  Muscle pain: Moderate | 11.6 [9.7 to 13.7]
  Muscle pain: Severe | 1.1 [0.5 to 1.9]
  Joint pain: Any | 19.6 [17.3 to 22.2]
  Joint pain: Mild | 10.2 [8.5 to 12.3]
  Joint pain: Moderate | 8.6 [7.0 to 10.5]
  Joint pain: Severe | 0.8 [0.3 to 1.5]

6. Primary Outcome: Stage1: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2 (Group 2 and 4 Combined)
Description: Systemic events fever, vomiting, diarrhea, headache, fatigue, chills, muscle pain other than muscle pain at the injection site, and joint pain were recorded by using an e-diary. Fever was defined as >=38.0 degree C and categorized to 38.0 to 38.4 degree C, 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and >40.0 degree C. Headache, fatigue, chills, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily activity). Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required IV hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 in 24 hours).
Time Frame: 7 days after Vaccination 2
Population: Vaccination 2 safety population included participants who received the second dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 3 (Month 6), and for whom safety information from Visit 3 (Month 6) up to and including Visit 4 (month 7) was available. Here, "Overall Number of Participants Analyzed": number of participants with known values. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 903
Percentage of participants
  Fever: >= 38.0 degree C | 3.2 [2.2 to 4.6]
  Fever: 38.0 to 38.4 degree C | 1.9 [1.1 to 3.0]
  Fever: 38.5 to 38.9 degree C | 0.7 [0.2 to 1.4]
  Fever: 39.0 to 40.0 degree C | 0.7 [0.2 to 1.4]
  Fever: > 40.0 degree C | 0.0 [0.0 to 0.4]
  Fatigue: Any | 45.2 [41.9 to 48.5]
  Fatigue: Mild | 23.0 [20.3 to 25.9]
  Fatigue: Moderate | 19.2 [16.6 to 21.9]
  Fatigue: Severe | 3.0 [2.0 to 4.3]
  Headache: Any | 41.6 [38.4 to 44.9]
  Headache: Mild | 23.1 [20.4 to 26.0]
  Headache: Moderate | 16.5 [14.1 to 19.1]
  Headache: Severe | 2.0 [1.2 to 3.1]
  Chills: Any | 18.5 [16.0 to 21.2]
  Chills: Mild | 11.6 [9.6 to 13.9]
  Chills: Moderate | 6.2 [4.7 to 8.0]
  Chills: Severe | 0.7 [0.2 to 1.4]
  Vomiting: Any | 2.8 [1.8 to 4.1]
  Vomiting: Mild | 2.0 [1.2 to 3.1]
  Vomiting: Moderate | 0.8 [0.3 to 1.6]
  Vomiting: Severe | 0.0 [0.0 to 0.4]
  Diarrhea: Any | 10.6 [8.7 to 12.8]
  Diarrhea: Mild | 7.6 [6.0 to 9.6]
  Diarrhea: Moderate | 2.5 [1.6 to 3.8]
  Diarrhea: Severe | 0.4 [0.1 to 1.1]
  Muscle pain: Any | 21.4 [18.7 to 24.2]
  Muscle pain: Mild | 11.5 [9.5 to 13.8]
  Muscle pain: Moderate | 7.8 [6.1 to 9.7]
  Muscle pain: Severe | 2.1 [1.3 to 3.3]
  Joint pain: Any | 18.7 [16.2 to 21.4]
  Joint pain: Mild | 11.2 [9.2 to 13.4]
  Joint pain: Moderate | 6.5 [5.0 to 8.3]
  Joint pain: Severe | 1.0 [0.5 to 1.9]

7. Primary Outcome: Stage1: Percentage of Participants With Antipyretic Medication Use Within 7 Days After Vaccination 1 (Group 2 and 4 Combined)
Time Frame: 7 days after Vaccination 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1044
Percentage of participants | 18.6 [16.3 to 21.1]

8. Primary Outcome: Stage1: Percentage of Participants With Antipyretic Medication Use Within 7 Days After Vaccination 2 (Group 2 and 4 Combined)
Time Frame: 7 days after Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 903
Percentage of participants | 14.4 [12.2 to 16.9]

9. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Vaccination 1 (Group 2 and 4 Combined)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. Or that was considered to be an important medical event.
Time Frame: 30 days after Vaccination 1
Population: Vaccination 1 safety population included participants who received the first dose of investigational product (MenABCWY+saline or bivalent rLP2086+MenACWY-CRM) at Visit 1 (Month 0), and for whom safety information from Visit 1 (Month 0) to prior to Visit 3 (Month 6) was available. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 0.0 [0.0 to 0.3]

10. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Vaccination 2 (Group 2 and 4 Combined)
Description: as for outcome 9
Time Frame: 30 days after Vaccination 2
Population: Vaccination 2 safety population included participants who received the second dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 3 (Month 6), and for whom safety information from Visit 3 (Month 6) up to and including Visit 4 (month 7) was available. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 946
Percentage of participants | 0.0 [0.0 to 0.4]

11. Primary Outcome: Stage1: Percentage of Participants With at Least 1 SAE Within 30 Days After Any Vaccination (Group 2 and 4 Combined)
Description: as for outcome 9
Time Frame: 30 days after any vaccination
Population: Stage 1 Safety population: participants who had received at least 1 dose of investigational product during Stage 1 and for whom safety data were available. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 0.0 [0.0 to 0.3]

12. Primary Outcome: Stage1: Percentage of Participants With at Least 1 SAE During the Stage 1 Vaccination Phase (Group 2 and 4 Combined)
Description: as for outcome 9
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 0.8 [0.3 to 1.5]

13. Primary Outcome: Stage1: Percentage of Participants With at Least 1 SAE During the Stage 1 Follow-up Phase (Group 2 and 4 Combined)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. Or that was considered to be an important medical event. There was one participant who did not meet criteria for Stage 1 follow-up safety population. The subject's SAE happened in the follow-up phase but was not included in the follow-up safety population for Stage 1 (but in the safety population for Stage 1). Therefore, the SAE was not included in the follow-up table but in the broadly defined throughout Stage 1 table.
Time Frame: Stage 1 Follow-up phase: From 1 month after Vaccination 2 through 6 months after Vaccination 2 (5 Months)
Population: Stage 1 Follow-up Safety population: participants who received at least 1 dose of investigational product and for whom safety information was available from after Visit 4 (Month 7) up to and including Visit 5 (Month 12). Analysis was planned for combined Group 2 and 4. Here overall number of participants analysed included those participants who met criteria for Stage 1 Follow-up safety population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 950
Percentage of participants | 0.5 [0.2 to 1.2]

14. Primary Outcome: Stage1: Percentage of Participants With at Least 1 SAE Throughout the Stage 1 (Group 2 and 4 Combined)
Description: as for outcome 13
Time Frame: Throughout Stage 1: From the Vaccination 1 through 6 months after Vaccination 2 (12 Months)
Population: Stage 1 Safety population: participants who had received at least 1 dose of investigational product during Stage 1 and for whom safety data were available. Analysis was planned for combined Group 2 and 4. Here overall number of participants analysed included those participants who met criteria for Stage 1 safety population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 1.3 [0.7 to 2.2]

15. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Vaccination 1 (Group 2 and 4 Combined)
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: 30 days after Vaccination 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 6.3 [4.9 to 8.0]

16. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Vaccination 2 (Group 2 and 4 Combined)
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: 30 days after Vaccination 2
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 946
Percentage of participants | 8.8 [7.0 to 10.8]

17. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Any Vaccination (Group 2 and 4 Combined)
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: 30 days after any vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 13.3 [11.3 to 15.5]

18. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE During the Stage 1 Vaccination Phase (Group 2 and 4 Combined)
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 26.7 [24.0 to 29.5]

19. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE During the Stage 1 Follow-up Phase (Group 2 and 4 Combined)
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Stage 1 Follow-up phase: From 1 month after Vaccination 2 through 6 months after Vaccination 2 (5 Months)
Population: Stage 1 Follow-up Safety population: participants who received at least 1 dose of investigational product and for whom safety information was available from after Visit 4 (Month 7) up to and including Visit 5 (Month 12). Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 950
Percentage of participants | 16.6 [14.3 to 19.2]

20. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE Throughout the Stage 1 (Group 2 and 4 Combined)
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Throughout Stage 1: From the Vaccination 1 through 6 months after Vaccination 2 (12 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 33.7 [30.8 to 36.6]

21. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition (NDCMC) Within 30 Days After Vaccination 1 (Group 2 and 4 Combined)
Description: A NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: 30 days after Vaccination 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 0.3 [0.1 to 0.8]

22. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition (NDCMC) Within 30 Days After Vaccination 2 (Group 2 and 4 Combined)
Description: as for outcome 21
Time Frame: 30 days after Vaccination 2
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 946
Percentage of participants | 0.2 [0.0 to 0.8]

23. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition (NDCMC) Within 30 Days After Any Vaccination (Group 2 and 4 Combined)
Description: as for outcome 21
Time Frame: 30 days after any Vaccination
Population: Safety population for Stage 1 included participants who had received at least 1 dose of investigational product during Stage 1 and for whom safety data were available. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 0.5 [0.2 to 1.1]

24. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition (NDCMC) During the Stage 1 Vaccination Phase (Group 2 and 4 Combined)
Description: as for outcome 21
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 0.8 [0.3 to 1.5]

25. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition (NDCMC) During the Stage 1 Follow-up Phase (Group 2 and 4 Combined)
Description: as for outcome 21
Time Frame: Stage 1 Follow-up phase: From 1 month after Vaccination 2 through 6 months after Vaccination 2 (5 Months)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 950
Percentage of participants | 0.3 [0.1 to 0.9]

26. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition (NDCMC) Throughout the Stage 1 (Group 2 and 4)
Description: as for outcome 21
Time Frame: Throughout Stage 1: From the Vaccination 1 through 6 months after Vaccination 2 (12 Months)
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 0.9 [0.5 to 1.7]

27. Primary Outcome: Stage1: Percentage of Participants With at Least 1 AE Within 30 Days After Vaccination 1 (Group 2 and 4 Combined)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs did not include local reaction and systemic events collected by systematic approach.
Time Frame: 30 days after Vaccination 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 13.8 [11.8 to 16.0]

28. Primary Outcome: Stage1: Percentage of Participants With at Least 1 AE Within 30 Days After Vaccination 2 (Group 2 and 4 Combined)
Description: as for outcome 27
Time Frame: 30 days after Vaccination 2
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 946
Percentage of participants | 14.7 [12.5 to 17.1]

29. Primary Outcome: Stage1: Percentage of Participants With at Least 1 AE Within 30 Days After Any Vaccination (Group 2 and 4 Combined)
Description: as for outcome 27
Time Frame: 30 days after any vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 24.1 [21.6 to 26.8]

30. Primary Outcome: Stage1: Percentage of Participants With at Least 1 AE During Vaccination Phase (Group 2 and 4 Combined)
Description: as for outcome 27
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 40.7 [37.7 to 43.7]

31. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Immediate AE After Vaccination 1 (Group 2 and 4 Combined)
Description: Immediate AE was defined as AE occurring within the first 30 minutes after investigational product administration.
Time Frame: 30 minutes after Vaccination 1
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Percentage of participants | 0.9 [0.4 to 1.6]

32. Primary Outcome: Stage1: Percentage of Participants With at Least 1 Immediate AE After Vaccination 2 (Group 2 and 4 Combined)
Description: Immediate AE was defined as AE occurring within the first 30 minutes after investigational product administration.
Time Frame: 30 minutes after Vaccination 2
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 946
Percentage of participants | 0.3 [0.1 to 0.9]

33. Primary Outcome: Stage1: Number of Participants Who Missed School/Work Due to AE During the Stage 1 Vaccination Phase (Group 2 and 4 Combined)
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 1057
Participants | 171

34. Primary Outcome: Stage2: Percentage of Participants With Local Reactions Within 7 Days After Booster Vaccination: Group 1 Through Group 4
Description: as for outcome 3
Time Frame: 7 days after booster vaccination
Population: Booster vaccination safety population included participants who received the booster dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 10 (Month 54), and for whom safety information from Visit 10 (Month 54) up to and including Visit 11 (Month 55) was available. Here, 'Overall Number of Participants Analyzed' signifies number of participants with known values.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 1: MenABCWY + Saline (ACWY-Naive): Stage 1: ACWY-naive participants were randomized to receive an intramuscular injection of 0.5 milliliter (mL) of Neisseria meningitidis groups A, B, C, W, and Y vaccine (MenABCWY) and 0.5 mL of saline at Month 0, participants received 0.5 mL of MenABCWY vaccine intramuscularly at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received 0.5 mL of MenABCWY vaccine (booster vaccination) intramuscularly at Month 54.
- Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive): Stage 1: ACWY-naive participants were randomized to receive an intramuscular injection of 0.5 mL bivalent recombinant lipoprotein 2086 (rLP2086) vaccine and 0.5 mL of meningococcal group A, C, W-135, and Y conjugate vaccine (MenACWY-CRM) at Month 0. Participants received 0.5 mL of bivalent rLP2086 vaccine at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received intramuscularly injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL of MenACWY-CRM vaccine (booster vaccination) at Month 54.
- Group 3: MenABCWY + Saline (ACWY-Experienced): Stage 1: ACWY-experienced participants were randomized to receive an intramuscular injection of 0.5 milliliter (mL) of Neisseria meningitidis groups A, B, C, W, and Y vaccine (MenABCWY) and 0.5 mL of saline at Month 0, Participants received 0.5 mL of MenABCWY vaccine intramuscularly at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received 0.5 mL of MenABCWY vaccine (booster vaccination) intramuscularly at Month 54.
- Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced): Stage 1: ACWY-experienced participants were randomized to receive an intramuscular injection of 0.5 mL bivalent recombinant lipoprotein 2086 (rLP2086) vaccine and 0.5 mL of meningococcal group A, C, W-135, and Y conjugate vaccine (MenACWY-CRM) at Month 0. Participants received 0.5 mL of bivalent rLP2086 vaccine at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received intramuscularly injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL of MenACWY-CRM vaccine (booster vaccination) at Month 54.
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 59 | 35 | 74 | 55
Percentage of participants
  Redness: Any | 13.6 [6.0 to 25.0] | 28.6 [14.6 to 46.3] | 21.6 [12.9 to 32.7] | 25.5 [14.7 to 39.0]
  Redness: Mild | 5.1 [1.1 to 14.1] | 11.4 [3.2 to 26.7] | 9.5 [3.9 to 18.5] | 14.5 [6.5 to 26.7]
  Redness: Moderate | 3.4 [0.4 to 11.7] | 11.4 [3.2 to 26.7] | 8.1 [3.0 to 16.8] | 9.1 [3.0 to 20.0]
  Redness: Severe | 5.1 [1.1 to 14.1] | 5.7 [0.7 to 19.2] | 4.1 [0.8 to 11.4] | 1.8 [0.0 to 9.7]
  Swelling: Any | 18.6 [9.7 to 30.9] | 25.7 [12.5 to 43.3] | 18.9 [10.7 to 29.7] | 18.2 [9.1 to 30.9]
  Swelling: Mild | 10.2 [3.8 to 20.8] | 11.4 [3.2 to 26.7] | 6.8 [2.2 to 15.1] | 9.1 [3.0 to 20.0]
  Swelling: Moderate | 8.5 [2.8 to 18.7] | 11.4 [3.2 to 26.7] | 12.2 [5.7 to 21.8] | 7.3 [2.0 to 17.6]
  Swelling: Severe | 0.0 [0.0 to 6.1] | 2.9 [0.1 to 14.9] | 0.0 [0.0 to 4.9] | 1.8 [0.0 to 9.7]
  Pain at injection site: Any: number analyzed (Participants) | 58 | 35 | 74 | 55
  Pain at injection site: Any | 79.3 [66.6 to 88.8] | 85.7 [69.7 to 95.2] | 85.1 [75.0 to 92.3] | 85.5 [73.3 to 93.5]
  Pain at injection site: Mild: number analyzed (Participants) | 58 | 35 | 74 | 55
  Pain at injection site: Mild | 41.4 [28.6 to 55.1] | 25.7 [12.5 to 43.3] | 36.5 [25.6 to 48.5] | 47.3 [33.7 to 61.2]
  Pain at injection site: Moderate: number analyzed (Participants) | 58 | 35 | 74 | 55
  Pain at injection site: Moderate | 36.2 [24.0 to 49.9] | 45.7 [28.8 to 63.4] | 47.3 [35.6 to 59.3] | 38.2 [25.4 to 52.3]
  Pain at injection site: Severe: number analyzed (Participants) | 58 | 35 | 74 | 55
  Pain at injection site: Severe | 1.7 [0.0 to 9.2] | 14.3 [4.8 to 30.3] | 1.4 [0.0 to 7.3] | 0.0 [0.0 to 6.5]

35. Primary Outcome: Stage2: Percentage of Participants With Systemic Events Within 7 Days After Booster Vaccination: Group 1 Through Group 4
Description: Systemic events fever, vomiting, diarrhea, headache, fatigue, chills, muscle pain and joint pain were recorded in an e-diary. Fever was defined as >=38.0 degree Celsius (C) and categorized to 38.0 to 38.4 degree C, 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and >40.0 degree C. Headache, fatigue, chills, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily activity). Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required IV hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 in 24 hours).
Time Frame: 7 days after booster vaccination
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 60 | 39 | 76 | 56
Percentage of participants
  Fever: >= 38.0 degree C | 5.0 [1.0 to 13.9] | 2.6 [0.1 to 13.5] | 0.0 [0.0 to 4.7] | 1.8 [0.0 to 9.6]
  Fever: 38.0 to 38.4 degree C | 1.7 [0.0 to 8.9] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 4.7] | 1.8 [0.0 to 9.6]
  Fever: 38.4 to 38.9 degree C | 0.0 [0.0 to 6.0] | 2.6 [0.1 to 13.5] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 6.4]
  Fever: 38.9 to 40.0 degree C | 3.3 [0.4 to 11.5] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 6.4]
  Fever: > 40.0 degree C | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 6.4]
  Fatigue: Any | 46.7 [33.7 to 60.0] | 61.5 [44.6 to 76.6] | 61.8 [50.0 to 72.8] | 66.1 [52.2 to 78.2]
  Fatigue: Mild | 25.0 [14.7 to 37.9] | 25.6 [13.0 to 42.1] | 50.0 [38.3 to 61.7] | 37.5 [24.9 to 51.5]
  Fatigue: Moderate | 21.7 [12.1 to 34.2] | 30.8 [17.0 to 47.6] | 10.5 [4.7 to 19.7] | 23.2 [13.0 to 36.4]
  Fatigue: Severe | 0.0 [0.0 to 6.0] | 5.1 [0.6 to 17.3] | 1.3 [0.0 to 7.1] | 5.4 [1.1 to 14.9]
  Headache: Any | 36.7 [24.6 to 50.1] | 53.8 [37.2 to 69.9] | 46.1 [34.5 to 57.9] | 55.4 [41.5 to 68.7]
  Headache: Mild | 25.0 [14.7 to 37.9] | 20.5 [9.3 to 36.5] | 34.2 [23.7 to 46.0] | 39.3 [26.5 to 53.2]
  Headache: Moderate | 8.3 [2.8 to 18.4] | 28.2 [15.0 to 44.9] | 10.5 [4.7 to 19.7] | 14.3 [6.4 to 26.2]
  Headache: Severe | 3.3 [0.4 to 11.5] | 5.1 [0.6 to 17.3] | 1.3 [0.0 to 7.1] | 1.8 [0.0 to 9.6]
  Chills: Any | 10.0 [3.8 to 20.5] | 17.9 [7.5 to 33.5] | 18.4 [10.5 to 29.0] | 14.3 [6.4 to 26.2]
  Chills: Mild | 10.0 [3.8 to 20.5] | 12.8 [4.3 to 27.4] | 15.8 [8.4 to 26.0] | 12.5 [5.2 to 24.1]
  Chills: Moderate | 0.0 [0.0 to 6.0] | 5.1 [0.6 to 17.3] | 2.6 [0.3 to 9.2] | 0.0 [0.0 to 6.4]
  Chills: Severe | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 4.7] | 1.8 [0.0 to 9.6]
  Vomiting: Any | 3.3 [0.4 to 11.5] | 0.0 [0.0 to 9.0] | 2.6 [0.3 to 9.2] | 1.8 [0.0 to 9.6]
  Vomiting: Mild | 1.7 [0.0 to 8.9] | 0.0 [0.0 to 9.0] | 1.3 [0.0 to 7.1] | 1.8 [0.0 to 9.6]
  Vomiting: Moderate | 1.7 [0.0 to 8.9] | 0.0 [0.0 to 9.0] | 1.3 [0.0 to 7.1] | 0.0 [0.0 to 6.4]
  Vomiting: severe | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 6.4]
  Diarrhea: Any | 5.0 [1.0 to 13.9] | 10.3 [2.9 to 24.2] | 9.2 [3.8 to 18.1] | 12.5 [5.2 to 24.1]
  Diarrhea: Mild | 5.0 [1.0 to 13.9] | 7.7 [1.6 to 20.9] | 7.9 [3.0 to 16.4] | 7.1 [2.0 to 17.3]
  Diarrhea: Moderate | 0.0 [0.0 to 6.0] | 2.6 [0.1 to 13.5] | 1.3 [0.0 to 7.1] | 5.4 [1.1 to 14.9]
  Diarrhea: Severe | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 6.4]
  Muscle Pain: Any | 18.3 [9.5 to 30.4] | 30.8 [17.0 to 47.6] | 31.6 [21.4 to 43.3] | 23.2 [13.0 to 36.4]
  Muscle pain: Mild | 13.3 [5.9 to 24.6] | 10.3 [2.9 to 24.2] | 22.4 [13.6 to 33.4] | 19.6 [10.2 to 32.4]
  Muscle pain: Moderate | 5.0 [1.0 to 13.9] | 12.8 [4.3 to 27.4] | 7.9 [3.0 to 16.4] | 3.6 [0.4 to 12.3]
  Muscle pain: Severe | 0.0 [0.0 to 6.0] | 7.7 [1.6 to 20.9] | 1.3 [0.0 to 7.1] | 0.0 [0.0 to 6.4]
  Joint Pain: Any | 18.3 [9.5 to 30.4] | 25.6 [13.0 to 42.1] | 21.1 [12.5 to 31.9] | 16.1 [7.6 to 28.3]
  Joint pain: Mild | 15.0 [7.1 to 26.6] | 12.8 [4.3 to 27.4] | 11.8 [5.6 to 21.3] | 12.5 [5.2 to 24.1]
  Joint pain: Moderate | 3.3 [0.4 to 11.5] | 10.3 [2.9 to 24.2] | 9.2 [3.8 to 18.1] | 3.6 [0.4 to 12.3]
  Joint pain: Severe | 0.0 [0.0 to 6.0] | 2.6 [0.1 to 13.5] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 6.4]

36. Primary Outcome: Stage2: Percentage of Participants With Antipyretic Medication Use Within 7 Days After Booster Vaccination: Group 1 Through Group 4
Time Frame: 7 days after booster vaccination
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 60 | 39 | 76 | 56
Percentage of participants | 16.7 [8.3 to 28.5] | 20.5 [9.3 to 36.5] | 13.2 [6.5 to 22.9] | 10.7 [4.0 to 21.9]

37. Primary Outcome: Stage2: Percentage of Participants With at Least 1 SAE During Booster Vaccination Phase: Group 1 Through Group 4
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. Or that was considered to be an important medical event. SAE of "pregnancy" for one participant during the booster vaccination phase was recorded erroneously and hence it was included in results of Group 4.
Time Frame: Booster vaccination phase: From booster vaccination through 1 month after booster vaccination
Population: Booster vaccination safety population included participants who received the booster dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 10 (Month 54), and for whom safety information from Visit 10 (Month 54) up to and including Visit 11 (Month 55) was available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 40 | 77 | 56
Percentage of participants | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 4.7] | 1.8 [0.0 to 9.6]

38. Primary Outcome: Stage2: Percentage of Participants With at Least 1 SAE During the Booster Follow-up Phase: Group 1 Through Group 4
Description: as for outcome 9
Time Frame: Booster follow-up phase: From 1 month after booster vaccination through 6 months after booster vaccination (up to 5 months)
Population: Booster Follow-up safety population for Stage 2 included participants who received the booster dose of investigational product and for whom safety information was available from after Visit 11 (Month 55) up to and including Visit 12 (Month 60).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 38 | 77 | 56
Percentage of participants | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 9.3] | 2.6 [0.3 to 9.1] | 0.0 [0.0 to 6.4]

39. Primary Outcome: Stage2: Percentage of Participants With at Least 1 SAE Throughout Booster Phase: Group 1 Through Group 4
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. Or that was considered to be an important medical event. SAE of "pregnancy" for one participant during the booster vaccination phase was recorded erroneously and hence it was reported in result of outcome measure 37 for Group 4. Subsequently correction was made by the trial site and not included in subsequent phase/results. Hence, that 1 participant is not included in results of Group 4 here.
Time Frame: Throughout Booster phase: From booster vaccination through 6 months after booster vaccination
Population: Booster safety population included participants who received the booster dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 10 (Month 54), and for whom safety information from Visit 10 (Month 54) up to and including Visit 12 (Month 60) was available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced): Stage 1: ACWY-experienced participants were randomized to receive an intramuscular injection of 0.5 mL bivalent recombinant lipoprotein 2086 (rLP2086) vaccine and 0.5 mL of meningococcal group A, C, W-135, and Y conjugate vaccine (MenACWY-CRM) at Month 0.Participants received 0.5 mL of bivalent rLP2086 vaccine at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received intramuscularly injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL of MenACWY-CRM vaccine (booster vaccination) at Month 54.
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 40 | 77 | 56
Percentage of participants | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 8.8] | 2.6 [0.3 to 9.1] | 0.0 [0.0 to 6.4]

40. Primary Outcome: Stage2: Percentage of Participants With at Least 1 Medically Attended AE During Booster Vaccination Phase: Group 1 Through Group 4
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Booster vaccination phase: From booster vaccination through 1 month after booster vaccination
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 40 | 77 | 56
Percentage of participants | 9.0 [3.4 to 18.5] | 5.0 [0.6 to 16.9] | 2.6 [0.3 to 9.1] | 7.1 [2.0 to 17.3]

41. Primary Outcome: Stage2: Percentage of Participants With at Least 1 Medically Attended AE During the Booster Follow-up Phase: Group 1 Through Group 4
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: as for outcome 38
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 38 | 77 | 56
Percentage of participants | 3.0 [0.4 to 10.4] | 13.2 [4.4 to 28.1] | 6.5 [2.1 to 14.5] | 7.1 [2.0 to 17.3]

42. Primary Outcome: Stage2: Percentage of Participants With at Least 1 Medically Attended AE Throughout Booster Phase: Group 1 Through Group 4
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Throughout Booster Phase: From booster vaccination through 6 months after booster vaccination
Population: as for outcome 39
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 40 | 77 | 56
Percentage of participants | 10.4 [4.3 to 20.3] | 15.0 [5.7 to 29.8] | 7.8 [2.9 to 16.2] | 14.3 [6.4 to 26.2]

43. Primary Outcome: Stage2: Percentage of Participants With at Least 1 NDCMC During Booster Vaccination Phase: Group 1 Through Group 4
Description: as for outcome 21
Time Frame: Booster Vaccination Phase: From booster vaccination through 1 month after booster vaccination
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 40 | 77 | 56
Percentage of participants | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 8.8] | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 6.4]

44. Primary Outcome: Stage2: Percentage of Participants With at Least 1 NDCMC During the Booster Follow-up Phase: Group 1 Through Group 4
Description: as for outcome 21
Time Frame: as for outcome 38
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 38 | 77 | 56
Percentage of participants | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 9.3] | 2.6 [0.3 to 9.1] | 0.0 [0.0 to 6.4]

45. Primary Outcome: Stage2: Percentage of Participants With at Least 1 NDCMC Throughout Booster Phase: Group 1 Through Group 4
Description: as for outcome 21
Time Frame: Throughout Booster Phase: From booster vaccination through 6 months after booster vaccination
Population: as for outcome 39
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 40 | 77 | 56
Percentage of participants | 0.0 [0.0 to 5.4] | 0.0 [0.0 to 8.8] | 2.6 [0.3 to 9.1] | 0.0 [0.0 to 6.4]

46. Primary Outcome: Stage2: Percentage of Participants With at Least 1 AE During Booster Vaccination Phase: Group 1 Through Group 4
Description: as for outcome 27
Time Frame: Booster Vaccination Phase: From booster vaccination through 1 month after booster vaccination
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 40 | 77 | 56
Percentage of participants | 13.4 [6.3 to 24.0] | 10.0 [2.8 to 23.7] | 10.4 [4.6 to 19.4] | 17.9 [8.9 to 30.4]

47. Primary Outcome: Stage2: Percentage of Participants With at Least 1 Immediate AE After Booster Vaccination: Group 1 Through Group 4
Description: Immediate AE was defined as AE occurring within the first 30 minutes after investigational product administration.
Time Frame: 30 minutes after booster vaccination
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 40 | 77 | 56
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

48. Primary Outcome: Stage2: Number of Participants Who Missed School/Work Due to AE After Booster Vaccination: Group 1 Through Group 4
Time Frame: Booster Vaccination Phase: From booster vaccination through 1 month after booster vaccination
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 67 | 40 | 77 | 56
Participants | 3 | 0 | 3 | 2

49. Secondary Outcome: Stage1: Percentage of Participants With hSBA Titer Level >= LLOQ for 4 Primary MenB Test Strains 1 Month After Vaccination 2 (Group 2 and 4 Combined)
Description: Percentage of participants who achieved an hSBA titer >= LLOQ for all 4 primary MenB test strains combined (LLOQ was 1:16 for A22 and 1:8 for A56, B24, and B44) was reported in this outcome measure. Four primary MenB test strains were PMB80 (A22), PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44).
Time Frame: 1 month after Vaccination 2
Population: Stage 1 EIP analyzed. Here "Overall Number of Participants analyzed" included all participants who were measured and analyzed. Here, 'Number Analyzed' signifies number of participants with valid and determinate hSBA results on all 4 strains at given time point. Analysis was planned combined for Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM): Stage 1: ACWY-naive and experienced participants who received an intramuscular injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL MenACWY-CRM vaccine at Month 0. Participants received 0.5 mL of bivalent rLP2086 vaccine at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received an intramuscular injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL MenACWY-CRM vaccine at Month 54.
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 864
Percentage of participants
  PMB80 (A22) 1 month after Vaccination 2: number analyzed (Participants) | 852
  PMB80 (A22) 1 month after Vaccination 2 | 91.0 [88.8 to 92.8]
  PMB2001 (A56) 1 month after Vaccination 2: number analyzed (Participants) | 854
  PMB2001 (A56) 1 month after Vaccination 2 | 99.4 [98.6 to 99.8]
  PMB2948 (B24) 1 month after Vaccination 2: number analyzed (Participants) | 842
  PMB2948 (B24) 1 month after Vaccination 2 | 79.3 [76.4 to 82.0]
  PMB2707 (B44) 1 month after Vaccination 2: number analyzed (Participants) | 853
  PMB2707 (B44) 1 month after Vaccination 2 | 94.5 [92.7 to 95.9]

50. Secondary Outcome: Stage1: Percentage of Participants With hSBA Titer Level >= 1:4, >= 1:8, >= 1:16, >= 1:32, >= 1:64, >= 1:128 for All 4 Primary MenB Test Strains 1 Month After Vaccination 2 (Group 2 and 4 Combined)
Description: Percentage of participants who achieved an hSBA titer >= 1:4, >= 1:8, >= 1:16, >= 1:32, >= 1:64, >= 1:128 for all 4 primary MenB test strains was reported in this outcome measure. Four primary MenB test strains were PMB80 (A22), PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44).
Time Frame: 1 month after Vaccination 2 (Vacc 2)
Population: Stage 1 EIP analyzed. Here "Overall Number of Participants analyzed" included all participants who were measured and analyzed. Here, 'Number Analyzed' signifies number of participants with valid and determinate hSBA results on all 4 strains at given time point. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 864
Percentage of participants
  PMB80 (A22) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 852
  PMB80 (A22) 1 Month after Vacc 2 >=1:4 | 91.7 [89.6 to 93.4]
  PMB80 (A22) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 852
  PMB80 (A22) 1 Month after Vacc 2 >=1:8 | 91.5 [89.5 to 93.3]
  PMB80 (A22) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 852
  PMB80 (A22) 1 Month after Vacc 2 >=1:16 | 91.0 [88.8 to 92.8]
  PMB80 (A22) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 852
  PMB80 (A22) 1 Month after Vacc 2 >=1:32 | 80.2 [77.3 to 82.8]
  PMB80 (A22) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 852
  PMB80 (A22) 1 Month after Vacc 2 >=1:64 | 54.9 [51.5 to 58.3]
  PMB80 (A22) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 852
  PMB80 (A22) 1 Month after Vacc 2 >=1:128 | 27.3 [24.4 to 30.5]
  PMB2001 (A56) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 854
  PMB2001 (A56) 1 Month after Vacc 2 >=1:4 | 99.5 [98.8 to 99.9]
  PMB2001 (A56) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 854
  PMB2001 (A56) 1 Month after Vacc 2 >=1:8 | 99.4 [98.6 to 99.8]
  PMB2001 (A56) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 854
  PMB2001 (A56) 1 Month after Vacc 2 >=1:16 | 99.1 [98.2 to 99.6]
  PMB2001 (A56) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 854
  PMB2001 (A56) 1 Month after Vacc 2 >=1:32 | 97.0 [95.6 to 98.0]
  PMB2001 (A56) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 854
  PMB2001 (A56) 1 Month after Vacc 2 >=1:64 | 87.7 [85.3 to 89.8]
  PMB2001 (A56) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 854
  PMB2001 (A56) 1 Month after Vacc 2 >=1:128 | 69.2 [66.0 to 72.3]
  PMB2948 (B24) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 842
  PMB2948 (B24) 1 Month after Vacc 2 >=1:4 | 81.2 [78.4 to 83.8]
  PMB2948 (B24) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 842
  PMB2948 (B24) 1 Month after Vacc 2 >=1:8 | 79.3 [76.4 to 82.0]
  PMB2948 (B24) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 842
  PMB2948 (B24) 1 Month after Vacc 2 >=1:16 | 74.0 [70.9 to 76.9]
  PMB2948 (B24) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 842
  PMB2948 (B24) 1 Month after Vacc 2 >=1:32 | 47.9 [44.4 to 51.3]
  PMB2948 (B24) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 842
  PMB2948 (B24) 1 Month after Vacc 2 >=1:64 | 24.9 [22.1 to 28.0]
  PMB2948 (B24) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 842
  PMB2948 (B24) 1 Month after Vacc 2 >=1:128 | 9.6 [7.7 to 11.8]
  PMB2707 (B44) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 853
  PMB2707 (B44) 1 Month after Vacc 2 >=1:4 | 96.2 [94.7 to 97.4]
  PMB2707 (B44) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 853
  PMB2707 (B44) 1 Month after Vacc 2 >=1:8 | 94.5 [92.7 to 95.9]
  PMB2707 (B44) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 853
  PMB2707 (B44) 1 Month after Vacc 2 >=1:16 | 89.0 [86.7 to 91.0]
  PMB2707 (B44) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 853
  PMB2707 (B44) 1 Month after Vacc 2 >=1:32 | 68.6 [65.3 to 71.7]
  PMB2707 (B44) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 853
  PMB2707 (B44) 1 Month after Vacc 2 >=1:64 | 41.0 [37.7 to 44.4]
  PMB2707 (B44) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 853
  PMB2707 (B44) 1 Month after Vacc 2 >=1:128 | 19.2 [16.6 to 22.0]

51. Secondary Outcome: Stage1: hSBA Geometric Mean Titers (GMTs) for All 4 Primary MenB Test Strains Combined 1 Month After Vaccination 2 (Group 2 and 4 Combined)
Description: GMTs were calculated using all participants with valid and determinate hSBA titers at the given time point. LLOQ = 1:16 for A22; 1:8 for A56, B24, and B44. Titers below the LLOQ were set to 0.5 * LLOQ for analysis. Four primary MenB test strains were PMB80 (A22), PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44).
Time Frame: 1 month after Vaccination 2 (Vacc 2)
Population: as for outcome 50
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 864
Titers
  PMB80 (A22) 1 month after Vacc 2: number analyzed (Participants) | 852
  PMB80 (A22) 1 month after Vacc 2 | 49.3 [46.2 to 52.6]
  PMB2001 (A56) 1 month after Vacc 2: number analyzed (Participants) | 854
  PMB2001 (A56) 1 month after Vacc 2 | 139.5 [130.6 to 149.1]
  PMB2948 (B24) 1 month after Vacc 2: number analyzed (Participants) | 842
  PMB2948 (B24) 1 month after Vacc 2 | 21.2 [19.6 to 22.9]
  PMB2707 (B44) 1 month after Vacc 2: number analyzed (Participants) | 853
  PMB2707 (B44) 1 month after Vacc 2 | 37.8 [35.1 to 40.8]

52. Secondary Outcome: Stage1: Percentage of Participants With hSBA Titer Level >= LLOQ for 10 Secondary MenB Test Strains 1 Month After Vaccination 2 (Group 2 and 4 Combined)
Description: Percentage of participants who achieved an hSBA titer greater than or equal to LLOQ for 10 Secondary MenB test strains combined (LLOQ = 1:16 for A06, A12, and A19; 1:8 for A07, A15, A29, B03, B09, B15, and B16) was reported in this outcome measure.
Time Frame: 1 month after Vaccination 2 (Vacc 2)
Population: Stage 1 EIP analyzed. Here "Overall Number of Participants analyzed" included all participants who were measured and analyzed. Here, 'Number Analyzed' signifies number of participants with valid and determinate hSBA results on all 10 strains at given time point. Analysis was planned for combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 180
Percentage of participants
  PMB3175 (A29) 1 month after Vacc 2: number analyzed (Participants) | 166
  PMB3175 (A29) 1 month after Vacc 2 | 95.2 [90.7 to 97.9]
  PMB3010 (A06) 1 month after Vacc 2: number analyzed (Participants) | 159
  PMB3010 (A06) 1 month after Vacc 2 | 89.3 [83.4 to 93.6]
  PMB824 (A12) 1 month after Vacc 2: number analyzed (Participants) | 157
  PMB824 (A12) 1 month after Vacc 2 | 83.4 [76.7 to 88.9]
  PMB3040 (A07) 1 month after Vacc 2: number analyzed (Participants) | 157
  PMB3040 (A07) 1 month after Vacc 2 | 96.8 [92.7 to 99.0]
  PMB1672 (A15) 1 month after Vacc 2: number analyzed (Participants) | 165
  PMB1672 (A15) 1 month after Vacc 2 | 89.1 [83.3 to 93.4]
  PMB1989 (A19) 1 month after Vacc 2: number analyzed (Participants) | 167
  PMB1989 (A19) 1 month after Vacc 2 | 90.4 [84.9 to 94.4]
  PMB648 (B16) 1 month after Vacc 2: number analyzed (Participants) | 164
  PMB648 (B16) 1 month after Vacc 2 | 77.4 [70.3 to 83.6]
  PMB866 (B09) 1 month after Vacc 2: number analyzed (Participants) | 166
  PMB866 (B09) 1 month after Vacc 2 | 71.1 [63.6 to 77.8]
  PMB1256 (B03) 1 month after Vacc 2: number analyzed (Participants) | 164
  PMB1256 (B03) 1 month after Vacc 2 | 74.4 [67.0 to 80.9]
  PMB431 (B15) 1 month after Vacc 2: number analyzed (Participants) | 167
  PMB431 (B15) 1 month after Vacc 2 | 85.0 [78.7 to 90.1]

53. Secondary Outcome: Stage1: Percentage of Participants With hSBA Titer Level >= 1:4, >= 1:8, >= 1:16, >= 1:32, >= 1:64, >= 1:128 for Each of the 10 Secondary MenB Test Strains 1 Month After Vaccination 2 (Group 2 and 4 Combined)
Description: Percentage of participants who achieved an hSBA titer >= 1:4, >= 1:8, >= 1:16, >= 1:32, >= 1:64, >= 1:128 for each of the 10 secondary MenB test strains was reported in this outcome measure. 10 secondary MenB test strains were PMB3175 (A29), PMB3010 (A06), PMB824 (A12), PMB3040 (A07), PMB1672 (A15), PMB1989 (A19), PMB648 (B16), PMB866 (B09), PMB1256 (B03) and PMB431 (B15).
Time Frame: 1 month after Vaccination 2 (Vacc 2)
Population: as for outcome 52
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 180
Percentage of participants
  PMB3175 (A29) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 166
  PMB3175 (A29) 1 Month after Vacc 2 >=1:4 | 95.8 [91.5 to 98.3]
  PMB3175 (A29) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 166
  PMB3175 (A29) 1 Month after Vacc 2 >=1:8 | 95.2 [90.7 to 97.9]
  PMB3175 (A29) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 166
  PMB3175 (A29) 1 Month after Vacc 2 >=1:16 | 92.2 [87.0 to 95.8]
  PMB3175 (A29) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 166
  PMB3175 (A29) 1 Month after Vacc 2 >=1:32 | 71.7 [64.2 to 78.4]
  PMB3175 (A29) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 166
  PMB3175 (A29) 1 Month after Vacc 2 >=1:64 | 38.0 [30.5 to 45.8]
  PMB3175 (A29) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 166
  PMB3175 (A29) 1 Month after Vacc 2 >=1:128 | 13.9 [9.0 to 20.1]
  PMB3010 (A06) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 159
  PMB3010 (A06) 1 Month after Vacc 2 >=1:4 | 89.9 [84.2 to 94.1]
  PMB3010 (A06) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 159
  PMB3010 (A06) 1 Month after Vacc 2 >=1:8 | 89.3 [83.4 to 93.6]
  PMB3010 (A06) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 159
  PMB3010 (A06) 1 Month after Vacc 2 >=1:16 | 89.3 [83.4 to 93.6]
  PMB3010 (A06) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 159
  PMB3010 (A06) 1 Month after Vacc 2 >=1:32 | 79.9 [72.8 to 85.8]
  PMB3010 (A06) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 159
  PMB3010 (A06) 1 Month after Vacc 2 >=1:64 | 54.7 [46.6 to 62.6]
  PMB3010 (A06) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 159
  PMB3010 (A06) 1 Month after Vacc 2 >=1:128 | 22.0 [15.8 to 29.3]
  PMB824 (A12) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 157
  PMB824 (A12) 1 Month after Vacc 2 >=1:4 | 89.2 [83.2 to 93.6]
  PMB824 (A12) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 157
  PMB824 (A12) 1 Month after Vacc 2 >=1:8 | 87.9 [81.7 to 92.6]
  PMB824 (A12) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 157
  PMB824 (A12) 1 Month after Vacc 2 >=1:16 | 83.4 [76.7 to 88.9]
  PMB824 (A12) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 157
  PMB824 (A12) 1 Month after Vacc 2 >=1:32 | 52.9 [44.8 to 60.9]
  PMB824 (A12) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 157
  PMB824 (A12) 1 Month after Vacc 2 >=1:64 | 18.5 [12.7 to 25.4]
  PMB824 (A12) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 157
  PMB824 (A12) 1 Month after Vacc 2 >=1:128 | 1.3 [0.2 to 4.5]
  PMB3040 (A07) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 157
  PMB3040 (A07) 1 Month after Vacc 2 >=1:4 | 96.8 [92.7 to 99.0]
  PMB3040 (A07) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 157
  PMB3040 (A07) 1 Month after Vacc 2 >=1:8 | 96.8 [92.7 to 99.0]
  PMB3040 (A07) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 157
  PMB3040 (A07) 1 Month after Vacc 2 >=1:16 | 96.8 [92.7 to 99.0]
  PMB3040 (A07) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 157
  PMB3040 (A07) 1 Month after Vacc 2 >=1:32 | 94.3 [89.4 to 97.3]
  PMB3040 (A07) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 157
  PMB3040 (A07) 1 Month after Vacc 2 >=1:64 | 68.8 [60.9 to 75.9]
  PMB3040 (A07) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 157
  PMB3040 (A07) 1 Month after Vacc 2 >=1:128 | 31.2 [24.1 to 39.1]
  PMB1672 (A15) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 165
  PMB1672 (A15) 1 Month after Vacc 2 >=1:4 | 89.1 [83.3 to 93.4]
  PMB1672 (A15) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 165
  PMB1672 (A15) 1 Month after Vacc 2 >=1:8 | 89.1 [83.3 to 93.4]
  PMB1672 (A15) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 165
  PMB1672 (A15) 1 Month after Vacc 2 >=1:16 | 87.3 [81.2 to 91.9]
  PMB1672 (A15) (n=165) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 165
  PMB1672 (A15) (n=165) 1 Month after Vacc 2 >=1:32 | 69.7 [62.1 to 76.6]
  PMB1672 (A15) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 165
  PMB1672 (A15) 1 Month after Vacc 2 >=1:64 | 30.3 [23.4 to 37.9]
  PMB1672 (A15) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 165
  PMB1672 (A15) 1 Month after Vacc 2 >=1:128 | 5.5 [2.5 to 10.1]
  PMB1989 (A19) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 167
  PMB1989 (A19) 1 Month after Vacc 2 >=1:4 | 92.2 [87.1 to 95.8]
  PMB1989 (A19) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 167
  PMB1989 (A19) 1 Month after Vacc 2 >=1:8 | 92.2 [87.1 to 95.8]
  PMB1989 (A19) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 167
  PMB1989 (A19) 1 Month after Vacc 2 >=1:16 | 90.4 [84.9 to 94.4]
  PMB1989 (A19) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 167
  PMB1989 (A19) 1 Month after Vacc 2 >=1:32 | 84.4 [78.0 to 89.6]
  PMB1989 (A19) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 167
  PMB1989 (A19) 1 Month after Vacc 2 >=1:64 | 61.1 [53.2 to 68.5]
  PMB1989 (A19) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 167
  PMB1989 (A19) 1 Month after Vacc 2 >=1:128 | 28.7 [22.0 to 36.2]
  PMB648 (B16) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 164
  PMB648 (B16) 1 Month after Vacc 2 >=1:4 | 79.3 [72.3 to 85.2]
  PMB648 (B16) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 164
  PMB648 (B16) 1 Month after Vacc 2 >=1:8 | 77.4 [70.3 to 83.6]
  PMB648 (B16) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 164
  PMB648 (B16) 1 Month after Vacc 2 >=1:16 | 73.8 [66.4 to 80.3]
  PMB648 (B16) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 164
  PMB648 (B16) 1 Month after Vacc 2 >=1:32 | 51.2 [43.3 to 59.1]
  PMB648 (B16) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 164
  PMB648 (B16) 1 Month after Vacc 2 >=1:64 | 28.7 [21.9 to 36.2]
  PMB648 (B16) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 164
  PMB648 (B16) 1 Month after Vacc 2 >=1:128 | 6.1 [3.0 to 10.9]
  PMB866 (B09) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 166
  PMB866 (B09) 1 Month after Vacc 2 >=1:4 | 74.7 [67.4 to 81.1]
  PMB866 (B09) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 166
  PMB866 (B09) 1 Month after Vacc 2 >=1:8 | 71.1 [63.6 to 77.8]
  PMB866 (B09) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 166
  PMB866 (B09) 1 Month after Vacc 2 >=1:16 | 63.3 [55.4 to 70.6]
  PMB866 (B09) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 166
  PMB866 (B09) 1 Month after Vacc 2 >=1:32 | 34.3 [27.2 to 42.1]
  PMB866 (B09) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 166
  PMB866 (B09) 1 Month after Vacc 2 >=1:64 | 8.4 [4.7 to 13.7]
  PMB866 (B09) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 166
  PMB866 (B09) 1 Month after Vacc 2 >=1:128 | 2.4 [0.7 to 6.1]
  PMB1256 (B03) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 164
  PMB1256 (B03) 1 Month after Vacc 2 >=1:4 | 77.4 [70.3 to 83.6]
  PMB1256 (B03) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 164
  PMB1256 (B03) 1 Month after Vacc 2 >=1:8 | 74.4 [67.0 to 80.9]
  PMB1256 (B03) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 164
  PMB1256 (B03) 1 Month after Vacc 2 >=1:16 | 64.0 [56.2 to 71.4]
  PMB1256 (B03) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 164
  PMB1256 (B03) 1 Month after Vacc 2 >=1:32 | 42.1 [34.4 to 50.0]
  PMB1256 (B03) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 164
  PMB1256 (B03) 1 Month after Vacc 2 >=1:64 | 23.2 [16.9 to 30.4]
  PMB1256 (B03) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 164
  PMB1256 (B03) 1 Month after Vacc 2 >=1:128 | 7.3 [3.8 to 12.4]
  PMB431 (B15) 1 Month after Vacc 2 >=1:4: number analyzed (Participants) | 167
  PMB431 (B15) 1 Month after Vacc 2 >=1:4 | 87.4 [81.4 to 92.0]
  PMB431 (B15) 1 Month after Vacc 2 >=1:8: number analyzed (Participants) | 167
  PMB431 (B15) 1 Month after Vacc 2 >=1:8 | 85.0 [78.7 to 90.1]
  PMB431 (B15) 1 Month after Vacc 2 >=1:16: number analyzed (Participants) | 167
  PMB431 (B15) 1 Month after Vacc 2 >=1:16 | 72.5 [65.0 to 79.1]
  PMB431 (B15) 1 Month after Vacc 2 >=1:32: number analyzed (Participants) | 167
  PMB431 (B15) 1 Month after Vacc 2 >=1:32 | 36.5 [29.2 to 44.3]
  PMB431 (B15) 1 Month after Vacc 2 >=1:64: number analyzed (Participants) | 167
  PMB431 (B15) 1 Month after Vacc 2 >=1:64 | 15.0 [9.9 to 21.3]
  PMB431 (B15) 1 Month after Vacc 2 >=1:128: number analyzed (Participants) | 167
  PMB431 (B15) 1 Month after Vacc 2 >=1:128 | 2.4 [0.7 to 6.0]

54. Secondary Outcome: Stage1: hSBA Geometric Mean Titers (GMTs) for Each of the 10 Secondary MenB Test Strains 1 Month After Vaccination 2 (Group 2 and 4 Combined)
Description: GMTs were calculated using all participants with valid and determinate hSBA titers at the given time point. LLOQ = 1:16 for A06, A12, and A19; 1:8 for A07, A15, A29, B03, B09, B15, and B16. Titers below the LLOQ were set to 0.5*LLOQ for analysis.
Time Frame: 1 month after Vaccination 2 (Vacc 2)
Population: as for outcome 52
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 180
Titers
  PMB3175 (A29) 1 month after Vacc 2: number analyzed (Participants) | 166
  PMB3175 (A29) 1 month after Vacc 2 | 35.7 [30.9 to 41.2]
  PMB3010 (A06) 1 month after Vacc 2: number analyzed (Participants) | 159
  PMB3010 (A06) 1 month after Vacc 2 | 46.0 [39.7 to 53.1]
  PMB824 (A12) 1 month after Vacc 2: number analyzed (Participants) | 157
  PMB824 (A12) 1 month after Vacc 2 | 23.7 [21.2 to 26.5]
  PMB3040 (A07) 1 month after Vacc 2: number analyzed (Participants) | 157
  PMB3040 (A07) 1 month after Vacc 2 | 60.7 [53.6 to 68.8]
  PMB1672 (A15) 1 month after Vacc 2: number analyzed (Participants) | 165
  PMB1672 (A15) 1 month after Vacc 2 | 28.4 [24.7 to 32.7]
  PMB1989 (A19) 1 month after Vacc 2: number analyzed (Participants) | 167
  PMB1989 (A19) 1 month after Vacc 2 | 53.5 [46.3 to 61.9]
  PMB648 (B16) 1 month after Vacc 2: number analyzed (Participants) | 164
  PMB648 (B16) 1 month after Vacc 2 | 20.8 [17.5 to 24.6]
  PMB866 (B09) 1 month after Vacc 2: number analyzed (Participants) | 166
  PMB866 (B09) 1 month after Vacc 2 | 13.9 [12.0 to 16.2]
  PMB1256 (B03) 1 month after Vacc 2: number analyzed (Participants) | 164
  PMB1256 (B03) 1 month after Vacc 2 | 17.7 [14.8 to 21.3]
  PMB431 (B15) 1 month after Vacc 2: number analyzed (Participants) | 167
  PMB431 (B15) 1 month after Vacc 2 | 17.3 [15.1 to 19.8]

55. Secondary Outcome: Stage1: Percentage of Participants With hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY Titers >=LLOQ for ACWY Test Strains 1 Month After the Vaccination 1: Groups 1, 2, 3 and 4
Description: Percentage of participants who achieved an hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY titer >=LLOQ for ACWY test strains (LLOQ = 1:8 for all MenA, MenC, MenW, and MenY strains) was reported in this outcome measure.
Time Frame: 1 month after Vaccination 1
Population: Stage 1 modified intent-to-treat (mITT) population: all randomized participants who had received at least 1 study vaccination, who had at least 1 valid and determinate primary strain MenB or MenA/C/W/Y assay result available at any time point from Month 0 to 7. "Overall Number of Participants Analyzed": participants who were measured and analyzed for the outcome measure. 'Number Analyzed': participants with valid and determinate hSBA results for ACWY test strains at the given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 272 | 534 | 271 | 523
Percentage of participants
  MenA: number analyzed (Participants) | 264 | 510 | 218 | 411
  MenA | 99.2 [97.3 to 99.9] | 98.4 [96.9 to 99.3] | 100.0 [98.3 to 100.0] | 99.3 [97.9 to 99.8]
  MenC: number analyzed (Participants) | 262 | 509 | 264 | 506
  MenC | 92.4 [88.5 to 95.3] | 88.6 [85.5 to 91.2] | 100.0 [98.6 to 100.0] | 99.4 [98.3 to 99.9]
  MenW: number analyzed (Participants) | 264 | 512 | 219 | 414
  MenW | 98.5 [96.2 to 99.6] | 95.5 [93.3 to 97.1] | 99.5 [97.5 to 100.0] | 99.5 [98.3 to 99.9]
  MenY: number analyzed (Participants) | 263 | 510 | 218 | 413
  MenY | 99.6 [97.9 to 100.0] | 96.9 [95.0 to 98.2] | 99.5 [97.5 to 100.0] | 99.8 [98.7 to 100.0]

56. Secondary Outcome: Stage1: Percentage of Participants With hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY Titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, and >=1:128 for ACWY Test Strains 1 Month After the Vaccination 1: Groups 1, 2, 3 and 4
Description: Percentage of participants who achieved an hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY titer >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, >=1:128 for ACWY test strains was reported in this outcome measure.
Time Frame: 1 month after Vaccination 1
Population: Stage 1 mITT population included all randomized participants who had received at least 1 study vaccination and who had at least 1 valid and determinate primary strain MenB or MenA/C/W/Y assay result available at any time point from 0 to 7 months. "Overall Number of Participants Analyzed": participants who were measured and analyzed for the outcome measure and 'Number Analyzed' signifies number of participants with valid and determinate hSBA results for ACWY test strains at the given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 272 | 534 | 271 | 523
Percentage of participants
  MenA >=1:4: number analyzed (Participants) | 264 | 510 | 218 | 411
  MenA >=1:4 | 99.6 [97.9 to 100.0] | 98.4 [96.9 to 99.3] | 100.0 [98.3 to 100.0] | 99.3 [97.9 to 99.8]
  MenA >=1:8: number analyzed (Participants) | 264 | 510 | 218 | 411
  MenA >=1:8 | 99.2 [97.3 to 99.9] | 98.4 [96.9 to 99.3] | 100.0 [98.3 to 100.0] | 99.3 [97.9 to 99.8]
  MenA >=1:16: number analyzed (Participants) | 264 | 510 | 218 | 411
  MenA >=1:16 | 98.5 [96.2 to 99.6] | 98.0 [96.4 to 99.1] | 100.0 [98.3 to 100.0] | 99.3 [97.9 to 99.8]
  MenA >=1:32: number analyzed (Participants) | 264 | 510 | 218 | 411
  MenA >=1:32 | 97.7 [95.1 to 99.2] | 93.9 [91.5 to 95.8] | 99.5 [97.5 to 100.0] | 99.0 [97.5 to 99.7]
  MenA >=1:64: number analyzed (Participants) | 264 | 510 | 218 | 411
  MenA >=1:64 | 90.9 [86.8 to 94.1] | 86.3 [83.0 to 89.1] | 99.1 [96.7 to 99.9] | 98.3 [96.5 to 99.3]
  MenA >= 1:128: number analyzed (Participants) | 264 | 510 | 218 | 411
  MenA >= 1:128 | 75.0 [69.3 to 80.1] | 71.2 [67.0 to 75.1] | 95.4 [91.7 to 97.8] | 96.4 [94.1 to 97.9]
  MenC >=1:4: number analyzed (Participants) | 262 | 509 | 264 | 506
  MenC >=1:4 | 95.4 [92.1 to 97.6] | 93.3 [90.8 to 95.3] | 100.0 [98.6 to 100.0] | 99.4 [98.3 to 99.9]
  MenC >=1:8: number analyzed (Participants) | 262 | 509 | 264 | 506
  MenC >=1:8 | 92.4 [88.5 to 95.3] | 88.6 [85.5 to 91.2] | 100.0 [98.6 to 100.0] | 99.4 [98.3 to 99.9]
  MenC >=1:16: number analyzed (Participants) | 262 | 509 | 264 | 506
  MenC >=1:16 | 88.2 [83.6 to 91.8] | 80.9 [77.3 to 84.3] | 100.0 [98.6 to 100.0] | 99.2 [98.0 to 99.8]
  MenC >=1:32: number analyzed (Participants) | 262 | 509 | 264 | 506
  MenC >=1:32 | 76.3 [70.7 to 81.3] | 67.8 [63.5 to 71.8] | 98.9 [96.7 to 99.8] | 98.2 [96.7 to 99.2]
  MenC >=1:64: number analyzed (Participants) | 262 | 509 | 264 | 506
  MenC >=1:64 | 61.8 [55.7 to 67.7] | 55.0 [50.6 to 59.4] | 97.3 [94.6 to 98.9] | 97.2 [95.4 to 98.5]
  MenC >=1:128: number analyzed (Participants) | 262 | 509 | 264 | 506
  MenC >=1:128 | 50.8 [44.5 to 57.0] | 45.6 [41.2 to 50.0] | 95.5 [92.2 to 97.6] | 94.1 [91.6 to 96.0]
  MenW >=1:4: number analyzed (Participants) | 264 | 512 | 219 | 414
  MenW >=1:4 | 99.6 [97.9 to 100.0] | 97.7 [95.9 to 98.8] | 100.0 [98.3 to 100.0] | 99.5 [98.3 to 99.9]
  MenW >=1:8: number analyzed (Participants) | 264 | 512 | 219 | 414
  MenW >=1:8 | 98.5 [96.2 to 99.6] | 95.5 [93.3 to 97.1] | 99.5 [97.5 to 100.0] | 99.5 [98.3 to 99.9]
  MenW >=1:16: number analyzed (Participants) | 264 | 512 | 219 | 414
  MenW >=1:16 | 96.2 [93.1 to 98.2] | 89.3 [86.2 to 91.8] | 99.5 [97.5 to 100.0] | 99.3 [97.9 to 99.9]
  MenW >=1:32: number analyzed (Participants) | 264 | 512 | 219 | 414
  MenW >=1:32 | 82.2 [77.0 to 86.6] | 75.0 [71.0 to 78.7] | 99.5 [97.5 to 100.0] | 98.1 [96.2 to 99.2]
  MenW >=1:64: number analyzed (Participants) | 264 | 512 | 219 | 414
  MenW >=1:64 | 65.9 [59.8 to 71.6] | 56.1 [51.6 to 60.4] | 99.1 [96.7 to 99.9] | 96.6 [94.4 to 98.1]
  MenW >=1:128: number analyzed (Participants) | 264 | 512 | 219 | 414
  MenW >=1:128 | 43.9 [37.9 to 50.2] | 38.1 [33.9 to 42.4] | 98.6 [96.0 to 99.7] | 94.0 [91.2 to 96.1]
  MenY >=1:4: number analyzed (Participants) | 263 | 510 | 218 | 413
  MenY >=1:4 | 100.0 [98.6 to 100.0] | 99.2 [98.0 to 99.8] | 99.5 [97.5 to 100.0] | 100.0 [99.1 to 100.0]
  MenY >=1:8: number analyzed (Participants) | 263 | 510 | 218 | 413
  MenY >=1:8 | 99.6 [97.9 to 100.0] | 96.9 [95.0 to 98.2] | 99.5 [97.5 to 100.0] | 99.8 [98.7 to 100.0]
  MenY >=1:16: number analyzed (Participants) | 263 | 510 | 218 | 413
  MenY >=1:16 | 98.9 [96.7 to 99.8] | 92.9 [90.4 to 95.0] | 99.5 [97.5 to 100.0] | 99.3 [97.9 to 99.8]
  MenY >=1:32: number analyzed (Participants) | 263 | 510 | 218 | 413
  MenY >=1:32 | 92.4 [88.5 to 95.3] | 82.4 [78.8 to 85.6] | 99.1 [96.7 to 99.9] | 99.0 [97.5 to 99.7]
  MenY >=1:64: number analyzed (Participants) | 263 | 510 | 218 | 413
  MenY >=1:64 | 78.3 [72.9 to 83.2] | 66.9 [62.6 to 70.9] | 99.1 [96.7 to 99.9] | 97.1 [95.0 to 98.5]
  MenY >=1:128: number analyzed (Participants) | 263 | 510 | 218 | 413
  MenY >=1:128 | 62.0 [55.8 to 67.9] | 48.6 [44.2 to 53.1] | 98.6 [96.0 to 99.7] | 94.9 [92.3 to 96.8]

57. Secondary Outcome: Stage1: hSBA Geometric Mean Titers (GMTs) for ACWY Test Strains 1 Month After Vaccination 1: Groups 1, 2, 3 and 4
Description: GMTs were calculated using all participants with valid and determinate hSBA titers at the given time point. LLOQ = 1:8 for all MenA, MenC, MenW, and MenY. Titers below the LLOQ were set to 0.5*LLOQ for analysis.
Time Frame: 1 month after Vaccination 1
Population: as for outcome 56
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 272 | 534 | 271 | 523
Titers
  MenA: number analyzed (Participants) | 264 | 510 | 218 | 411
  MenA | 215.8 [184.6 to 252.4] | 203.2 [178.7 to 231.0] | 568.6 [492.9 to 656.0] | 916.1 [809.1 to 1037.3]
  MenC: number analyzed (Participants) | 262 | 509 | 264 | 506
  MenC | 111.5 [87.2 to 142.6] | 81.4 [68.1 to 97.4] | 814.9 [689.4 to 963.2] | 827.0 [722.5 to 946.6]
  MenW: number analyzed (Participants) | 264 | 512 | 219 | 414
  MenW | 98.4 [80.7 to 120.0] | 71.2 [61.5 to 82.4] | 1214.9 [1032.0 to 1430.1] | 1176.7 [1017.9 to 1360.2]
  MenY: number analyzed (Participants) | 263 | 510 | 218 | 413
  MenY | 141.9 [118.8 to 169.4] | 96.6 [83.9 to 111.2] | 1174.0 [990.3 to 1391.9] | 1000.2 [872.1 to 1147.1]

58. Secondary Outcome: Stage1: Percentage of Participants With hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY Titers >=1:8 (or LLOQ, Whichever is Higher) for ACWY Test Strains 1 Month After the Vaccination 1 in Groups 2 and 4, and 1 Month After Vaccination 2 in Groups 1 and 3
Description: Percentage of participants who achieved an hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY titer >= LLOQ for ACWY test strains (LLOQ = 1:8 for all MenA, MenC, MenW, and MenY strains) was reported in this outcome measure.
Time Frame: For Group 2 and 4: 1 month after Vaccination 1; For Group 1 and 3: 1 month after Vaccination 2
Population: as for outcome 56
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced) | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 534 | 523 | 242 | 244
Percentage of participants
  MenA: number analyzed (Participants) | 510 | 411 | 232 | 191
  MenA | 98.4 [96.9 to 99.3] | 99.3 [97.9 to 99.8] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenC: number analyzed (Participants) | 509 | 506 | 231 | 237
  MenC | 88.6 [85.5 to 91.2] | 99.4 [98.3 to 99.9] | 100.0 [98.4 to 100.0] | 99.6 [97.7 to 100.0]
  MenW: number analyzed (Participants) | 512 | 414 | 233 | 191
  MenW | 95.5 [93.3 to 97.1] | 99.5 [98.3 to 99.9] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenY: number analyzed (Participants) | 510 | 413 | 233 | 191
  MenY | 96.9 [95.0 to 98.2] | 99.8 [98.7 to 100.0] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]

59. Secondary Outcome: Stage1: Percentage of Participants With MenA, MenC, MenW, and MenY Titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, and, >=1:128 for ACWY Test Strains 1 Month After Vaccination 1 in Groups 2 and 4, and 1 Month After Vaccination 2 in Groups 1 and 3
Description: as for outcome 56
Time Frame: For Group 2 and 4: 1 month after Vaccination 1; For Group 1 and 3: 1 month after Vaccination 2
Population: as for outcome 56
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced) | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 534 | 523 | 242 | 244
Percentage of participants
  MenA >=1:4: number analyzed (Participants) | 510 | 411 | 232 | 191
  MenA >=1:4 | 98.4 [96.9 to 99.3] | 99.3 [97.9 to 99.8] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenA >=1:8: number analyzed (Participants) | 510 | 411 | 232 | 191
  MenA >=1:8 | 98.4 [96.9 to 99.3] | 99.3 [97.9 to 99.8] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenA >=1:16: number analyzed (Participants) | 510 | 411 | 232 | 191
  MenA >=1:16 | 98.0 [96.4 to 99.1] | 99.3 [97.9 to 99.8] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenA >=1:32: number analyzed (Participants) | 510 | 411 | 232 | 191
  MenA >=1:32 | 93.9 [91.5 to 95.8] | 99.0 [97.5 to 99.7] | 97.8 [95.0 to 99.3] | 99.5 [97.1 to 100.0]
  MenA >=1:64: number analyzed (Participants) | 510 | 411 | 232 | 191
  MenA >=1:64 | 86.3 [83.0 to 89.1] | 98.3 [96.5 to 99.3] | 92.2 [88.0 to 95.3] | 97.4 [94.0 to 99.1]
  MenA >=1:128: number analyzed (Participants) | 510 | 411 | 232 | 191
  MenA >=1:128 | 71.2 [67.0 to 75.1] | 96.4 [94.1 to 97.9] | 69.4 [63.0 to 75.3] | 92.7 [88.0 to 95.9]
  MenC >=1:4: number analyzed (Participants) | 509 | 506 | 231 | 237
  MenC >=1:4 | 93.3 [90.8 to 95.3] | 99.4 [98.3 to 99.9] | 100.0 [98.4 to 100.0] | 99.6 [97.7 to 100.0]
  MenC >=1:8: number analyzed (Participants) | 509 | 506 | 231 | 237
  MenC >=1:8 | 88.6 [85.5 to 91.2] | 99.4 [98.3 to 99.9] | 100.0 [98.4 to 100.0] | 99.6 [97.7 to 100.0]
  MenC >=1:16: number analyzed (Participants) | 509 | 506 | 231 | 237
  MenC >=1:16 | 80.9 [77.3 to 84.3] | 99.2 [98.0 to 99.8] | 99.6 [97.6 to 100.0] | 99.6 [97.7 to 100.0]
  MenC >=1:32: number analyzed (Participants) | 509 | 506 | 231 | 237
  MenC >=1:32 | 67.8 [63.5 to 71.8] | 98.2 [96.7 to 99.2] | 97.4 [94.4 to 99.0] | 99.6 [97.7 to 100.0]
  MenC >=1:64: number analyzed (Participants) | 509 | 506 | 231 | 237
  MenC >=1:64 | 55.0 [50.6 to 59.4] | 97.2 [95.4 to 98.5] | 90.9 [86.4 to 94.3] | 98.3 [95.7 to 99.5]
  MenC >=1:128: number analyzed (Participants) | 509 | 506 | 231 | 237
  MenC >=1:128 | 45.6 [41.2 to 50.0] | 94.1 [91.6 to 96.0] | 78.8 [72.9 to 83.9] | 92.8 [88.8 to 95.8]
  MenW >=1:4: number analyzed (Participants) | 512 | 414 | 233 | 191
  MenW >=1:4 | 97.7 [95.9 to 98.8] | 99.5 [98.3 to 99.9] | 100.0 [98.4 to 100.0] | 100.0 [98.1 to 100.0]
  MenW >=1:8: number analyzed (Participants) | 512 | 414 | 233 | 191
  MenW >=1:8 | 95.5 [93.3 to 97.1] | 99.5 [98.3 to 99.9] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenW >=1:16: number analyzed (Participants) | 512 | 414 | 233 | 191
  MenW >=1:16 | 89.3 [86.2 to 91.8] | 99.3 [97.9 to 99.9] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenW >=1:32: number analyzed (Participants) | 512 | 414 | 233 | 191
  MenW >=1:32 | 75.0 [71.0 to 78.7] | 98.1 [96.2 to 99.2] | 99.6 [97.6 to 100.0] | 99.5 [97.1 to 100.0]
  MenW >=1:64: number analyzed (Participants) | 512 | 414 | 233 | 191
  MenW >=1:64 | 56.1 [51.6 to 60.4] | 96.6 [94.4 to 98.1] | 97.0 [93.9 to 98.8] | 99.0 [96.3 to 99.9]
  MenW >=1:128: number analyzed (Participants) | 512 | 414 | 233 | 191
  MenW >=1:128 | 38.1 [33.9 to 42.4] | 94.0 [91.2 to 96.1] | 89.7 [85.1 to 93.3] | 97.9 [94.7 to 99.4]
  MenY >=1:4: number analyzed (Participants) | 510 | 413 | 233 | 191
  MenY >=1:4 | 99.2 [98.0 to 99.8] | 100.0 [99.1 to 100.0] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenY >=1:8: number analyzed (Participants) | 510 | 413 | 233 | 191
  MenY >=1:8 | 96.9 [95.0 to 98.2] | 99.8 [98.7 to 100.0] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenY >=1:16: number analyzed (Participants) | 510 | 413 | 233 | 191
  MenY >=1:16 | 92.9 [90.4 to 95.0] | 99.3 [97.9 to 99.8] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenY >=1:32: number analyzed (Participants) | 510 | 413 | 233 | 191
  MenY >=1:32 | 82.4 [78.8 to 85.6] | 99.0 [97.5 to 99.7] | 100.0 [98.4 to 100.0] | 99.5 [97.1 to 100.0]
  MenY >=1:64: number analyzed (Participants) | 510 | 413 | 233 | 191
  MenY >=1:64 | 66.9 [62.6 to 70.9] | 97.1 [95.0 to 98.5] | 97.4 [94.5 to 99.0] | 99.5 [97.1 to 100.0]
  MenY >=1:128: number analyzed (Participants) | 510 | 413 | 233 | 191
  MenY >=1:128 | 48.6 [44.2 to 53.1] | 94.9 [92.3 to 96.8] | 89.7 [85.1 to 93.3] | 95.3 [91.2 to 97.8]

60. Secondary Outcome: Stage1: hSBA GMTs for ACWY Test Strains 1 Month After Vaccination 1 in Groups 2 and 4 and 1 Month After Vaccination 2 in Groups 1 and 3
Description: as for outcome 57
Time Frame: For Group 2 and 4: 1 month after Vaccination 1; For Group 1 and 3: 1 month after Vaccination 2
Population: as for outcome 56
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced) | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 534 | 523 | 242 | 244
Titers
  MenA: number analyzed (Participants) | 510 | 411 | 232 | 191
  MenA | 203.2 [178.7 to 231.0] | 916.1 [809.1 to 1037.3] | 151.3 [134.1 to 170.7] | 337.3 [291.7 to 390.0]
  MenC: number analyzed (Participants) | 509 | 506 | 231 | 237
  MenC | 81.4 [68.1 to 97.4] | 827.0 [722.5 to 946.6] | 229.1 [194.7 to 269.5] | 498.7 [429.1 to 579.6]
  MenW: number analyzed (Participants) | 512 | 414 | 233 | 191
  MenW | 71.2 [61.5 to 82.4] | 1176.7 [1017.9 to 1360.2] | 274.1 [242.7 to 309.7] | 570.9 [484.3 to 673.0]
  MenY: number analyzed (Participants) | 510 | 413 | 233 | 191
  MenY | 96.6 [83.9 to 111.2] | 1000.2 [872.1 to 1147.1] | 301.5 [266.6 to 341.0] | 558.6 [470.0 to 663.9]

61. Secondary Outcome: Stage1: Percentage of Participants With hSBA Titer Level >= LLOQ for 4 Primary MenB Test Strains 1 Month After Vaccination 2 (Group 1 and 3 Combined; Group 2 and 4 Combined)
Description: Percentage of participants who achieved an hSBA titer >=LLOQ for all 4 primary MenB test strains (LLOQ was 1:16 for A22 and 1:8 for A56, B24, and B44) was reported in this outcome measure.
Time Frame: 1 month after Vaccination 2 (Vacc 2)
Population: Stage 1 EIP analyzed. Here, "Overall Number of Participants Analyzed" signifies number of participants measured and analyzed for this outcome measure. "Number Analyzed" signifies number of participants with valid and determinate hSBA results for each strains at given time point. Analysis was planned for combined Group 1 and 3 and combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 1+3 Combined (MenABCWY + Saline): Stage 1: ACWY-naive and experienced participants who received an intramuscular injection of 0.5 mL of MenABCWY vaccine and 0.5 mL of saline at Month 0, participants received 0.5 mL of MenABCWY vaccine intramuscularly at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received 0.5 mL of MenABCWY vaccine (booster vaccination) intramuscularly at Month 54
Arm/Group | Group 1+3 Combined (MenABCWY + Saline) | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 438 | 864
Percentage of participants
  PMB80 (A22) 1 month after Vacc 2: number analyzed (Participants) | 433 | 852
  PMB80 (A22) 1 month after Vacc 2 | 91.0 [87.9 to 93.5] | 91.0 [88.8 to 92.8]
  PMB2001 (A56) 1 month after Vacc 2: number analyzed (Participants) | 435 | 854
  PMB2001 (A56) 1 month after Vacc 2 | 98.6 [97.0 to 99.5] | 99.4 [98.6 to 99.8]
  PMB2948 (B24) 1 month after Vacc 2: number analyzed (Participants) | 426 | 842
  PMB2948 (B24) 1 month after Vacc 2 | 84.3 [80.5 to 87.6] | 79.3 [76.4 to 82.0]
  PMB2707 (B44) 1 month after Vacc 2: number analyzed (Participants) | 436 | 853
  PMB2707 (B44) 1 month after Vacc 2 | 95.4 [93.0 to 97.2] | 94.5 [92.7 to 95.9]

62. Secondary Outcome: Stage1: Percentage of Participants With >=4 Fold Rise in hSBA for 4 Primary MenB Strains and Composite Response (hSBA >=LLOQ for All 4 Primary MenB Strains Combined) From Baseline-1 Month After Vaccination 2 (Group 1 and 3 Combined;Group 2 and 4 Combined)
Description: Percentage of participants who achieved an hSBA titer greater than or equal to LLOQ for all 4 primary MenB test strains combined (LLOQ was 1:16 for A22 and 1:8 for A56, B24, and B44) was reported in this outcome measure.
Time Frame: Baseline to 1 month after Vaccination 2
Population: Stage 1 EIP analyzed. Here, "Overall Number of Participants Analyzed" signifies number of participants measure and analyzed for this outcome measure. "Number Analyzed" signifies number of participants with valid and determinate hSBA results on all 4 strains at given time point. Analysis was planned for combined Group 1 and 3 and combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1+3 Combined (MenABCWY + Saline) | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 438 | 864
Percentage of participants
  PMB80 (A22): number analyzed (Participants) | 422 | 827
  PMB80 (A22) | 75.8 [71.5 to 79.8] | 73.8 [70.6 to 76.7]
  PMB2001 (A56): number analyzed (Participants) | 418 | 823
  PMB2001 (A56) | 94.7 [92.1 to 96.7] | 95.0 [93.3 to 96.4]
  PMB2948 (B24): number analyzed (Participants) | 422 | 835
  PMB2948 (B24) | 76.1 [71.7 to 80.1] | 67.4 [64.1 to 70.6]
  PMB2707 (B44): number analyzed (Participants) | 432 | 850
  PMB2707 (B44) | 91.7 [88.6 to 94.1] | 86.4 [83.9 to 88.6]
  Composite hSBA response: number analyzed (Participants) | 418 | 814
  Composite hSBA response | 79.9 [75.7 to 83.6] | 74.3 [71.2 to 77.3]

63. Secondary Outcome: Stage1: Percentage of Participants With hSBA Titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, and >=1:128 for Each of the 4 Primary MenB Test Strains From 1 Month After Vaccination 2 (Group 1 and 3 Combined; Group 2 and 4 Combined)
Description: Percentage of participants who achieved an hSBA titer >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, and >=1:128 for all 4 primary MenB test strains was reported in this outcome measure.
Time Frame: 1 month after Vaccination 2
Population: as for outcome 62
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1+3 Combined (MenABCWY + Saline) | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 438 | 864
Percentage of participants
  PMB80 (A22) >=1:4: number analyzed (Participants) | 433 | 852
  PMB80 (A22) >=1:4 | 91.9 [88.9 to 94.3] | 91.7 [89.6 to 93.4]
  PMB80 (A22) >=1:8: number analyzed (Participants) | 433 | 852
  PMB80 (A22) >=1:8 | 91.7 [88.7 to 94.1] | 91.5 [89.5 to 93.3]
  PMB80 (A22) >=1:16: number analyzed (Participants) | 433 | 852
  PMB80 (A22) >=1:16 | 91.0 [87.9 to 93.5] | 91.0 [88.8 to 92.8]
  PMB80 (A22) >=1:32: number analyzed (Participants) | 433 | 852
  PMB80 (A22) >=1:32 | 82.4 [78.5 to 85.9] | 80.2 [77.3 to 82.8]
  PMB80 (A22) >=1:64: number analyzed (Participants) | 433 | 852
  PMB80 (A22) >=1:64 | 58.0 [53.2 to 62.7] | 54.9 [51.5 to 58.3]
  PMB80 (A22) >=1:128: number analyzed (Participants) | 433 | 852
  PMB80 (A22) >=1:128 | 27.9 [23.8 to 32.4] | 27.3 [24.4 to 30.5]
  PMB2001 (A56) >=1:4: number analyzed (Participants) | 435 | 854
  PMB2001 (A56) >=1:4 | 98.9 [97.3 to 99.6] | 99.5 [98.8 to 99.9]
  PMB2001 (A56) >=1:8: number analyzed (Participants) | 435 | 854
  PMB2001 (A56) >=1:8 | 98.6 [97.0 to 99.5] | 99.4 [98.6 to 99.8]
  PMB2001 (A56) >=1:16: number analyzed (Participants) | 435 | 854
  PMB2001 (A56) >=1:16 | 98.6 [97.0 to 99.5] | 99.1 [98.2 to 99.6]
  PMB2001 (A56) >=1:32: number analyzed (Participants) | 435 | 854
  PMB2001 (A56) >=1:32 | 96.8 [94.7 to 98.2] | 97.0 [95.6 to 98.0]
  PMB2001 (A56) >=1:64: number analyzed (Participants) | 435 | 854
  PMB2001 (A56) >=1:64 | 90.1 [86.9 to 92.8] | 87.7 [85.3 to 89.8]
  PMB2001 (A56) >=1:128: number analyzed (Participants) | 435 | 854
  PMB2001 (A56) >=1:128 | 74.0 [69.6 to 78.1] | 69.2 [66.0 to 72.3]
  PMB2948 (B24) >=1:4: number analyzed (Participants) | 426 | 842
  PMB2948 (B24) >=1:4 | 86.9 [83.3 to 89.9] | 81.2 [78.4 to 83.8]
  PMB2948 (B24) >=1:8: number analyzed (Participants) | 426 | 842
  PMB2948 (B24) >=1:8 | 84.3 [80.5 to 87.6] | 79.3 [76.4 to 82.0]
  PMB2948 (B24) >=1:16: number analyzed (Participants) | 426 | 842
  PMB2948 (B24) >=1:16 | 80.8 [76.7 to 84.4] | 74.0 [70.9 to 76.9]
  PMB2948 (B24) >=1:32: number analyzed (Participants) | 426 | 842
  PMB2948 (B24) >=1:32 | 58.5 [53.6 to 63.2] | 47.9 [44.4 to 51.3]
  PMB2948 (B24) >=1:64: number analyzed (Participants) | 426 | 842
  PMB2948 (B24) >=1:64 | 31.0 [26.6 to 35.6] | 24.9 [22.1 to 28.0]
  PMB2948 (B24) >=1:128: number analyzed (Participants) | 426 | 842
  PMB2948 (B24) >=1:128 | 13.4 [10.3 to 17.0] | 9.6 [7.7 to 11.8]
  PMB2707 (B44) >=1:4: number analyzed (Participants) | 436 | 853
  PMB2707 (B44) >=1:4 | 97.2 [95.2 to 98.6] | 96.2 [94.7 to 97.4]
  PMB2707 (B44) >=1:8: number analyzed (Participants) | 436 | 853
  PMB2707 (B44) >=1:8 | 95.4 [93.0 to 97.2] | 94.5 [92.7 to 95.9]
  PMB2707 (B44) >=1:16: number analyzed (Participants) | 436 | 853
  PMB2707 (B44) >=1:16 | 92.4 [89.5 to 94.7] | 89.0 [86.7 to 91.0]
  PMB2707 (B44) >=1:32: number analyzed (Participants) | 436 | 853
  PMB2707 (B44) >=1:32 | 72.9 [68.5 to 77.1] | 68.6 [65.3 to 71.7]
  PMB2707 (B44) >=1:64: number analyzed (Participants) | 436 | 853
  PMB2707 (B44) >=1:64 | 48.9 [44.1 to 53.7] | 41.0 [37.7 to 44.4]
  PMB2707 (B44) >=1:128: number analyzed (Participants) | 436 | 853
  PMB2707 (B44) >=1:128 | 22.0 [18.2 to 26.2] | 19.2 [16.6 to 22.0]

64. Secondary Outcome: Stage1: hSBA GMTs for Each of the 4 Primary MenB Test Strains 1 Month After Vaccination 2 (Group 1 and 3 Combined; Group 2 and 4 Combined)
Description: GMTs were calculated using all participants with valid and determinate hSBA titers at the given time point. LLOQ =1:16 for A22; 1:8 for A56, B24, and B44. Titers below the LLOQ were set to 0.5*LLOQ for analysis.
Time Frame: 1 month after Vaccination 2
Population: as for outcome 62
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1+3 Combined (MenABCWY + Saline) | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 438 | 864
Titers
  PMB80 (A22): number analyzed (Participants) | 433 | 852
  PMB80 (A22) | 51.0 [46.7 to 55.7] | 49.3 [46.2 to 52.6]
  PMB2001 (A56): number analyzed (Participants) | 435 | 854
  PMB2001 (A56) | 152.3 [138.5 to 167.5] | 139.5 [130.6 to 149.1]
  PMB2948 (B24): number analyzed (Participants) | 426 | 842
  PMB2948 (B24) | 26.6 [23.9 to 29.7] | 21.2 [19.6 to 22.9]
  PMB2707 (B44): number analyzed (Participants) | 436 | 853
  PMB2707 (B44) | 43.3 [39.1 to 47.9] | 37.8 [35.1 to 40.8]

65. Secondary Outcome: Stage1: Percentage of Participants With hSBA-MenA, hSBA-MenC, hSBA-MenW and hSBA-MenY Titers >=1:8 (or LLOQ) for ACWY Test Strains Before Vaccination 1 and Before Vaccination 2: Groups 1, 2, 3 and 4
Description: as for outcome 55
Time Frame: Before Vaccination 1 (Vacc 1) [Day 1], Before Vaccination 2 (Vacc 2) [173 to 194 Days After Visit 1]
Population: as for outcome 56
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 272 | 534 | 271 | 523
Percentage of participants
  MenA Before Vacc 1: number analyzed (Participants) | 270 | 528 | 219 | 418
  MenA Before Vacc 1 | 15.9 [11.8 to 20.8] | 22.9 [19.4 to 26.7] | 53.9 [47.0 to 60.6] | 52.6 [47.7 to 57.5]
  MenA Before Vacc 2: number analyzed (Participants) | 238 | 463 | 200 | 385
  MenA Before Vacc 2 | 91.6 [87.3 to 94.8] | 86.2 [82.7 to 89.2] | 99.0 [96.4 to 99.9] | 98.4 [96.6 to 99.4]
  MenC Before Vacc 1: number analyzed (Participants) | 267 | 526 | 264 | 511
  MenC Before Vacc 1 | 38.6 [32.7 to 44.7] | 39.0 [34.8 to 43.3] | 59.5 [53.3 to 65.4] | 61.1 [56.7 to 65.3]
  MenC Before Vacc 2: number analyzed (Participants) | 239 | 460 | 243 | 474
  MenC Before Vacc 2 | 92.9 [88.9 to 95.8] | 76.5 [72.4 to 80.3] | 98.4 [95.8 to 99.5] | 98.3 [96.7 to 99.3]
  MenW Before Vacc 1: number analyzed (Participants) | 268 | 527 | 218 | 418
  MenW Before Vacc 1 | 32.1 [26.5 to 38.0] | 34.5 [30.5 to 38.8] | 61.9 [55.1 to 68.4] | 60.8 [55.9 to 65.5]
  MenW Before Vacc 2: number analyzed (Participants) | 242 | 467 | 199 | 385
  MenW Before Vacc 2 | 99.2 [97.0 to 99.9] | 91.0 [88.0 to 93.4] | 100.0 [98.2 to 100.0] | 99.0 [97.4 to 99.7]
  MenY Before Vacc 1: number analyzed (Participants) | 265 | 528 | 219 | 421
  MenY Before Vacc 1 | 54.0 [47.8 to 60.1] | 58.1 [53.8 to 62.4] | 79.9 [74.0 to 85.0] | 77.9 [73.6 to 81.8]
  MenY Before Vacc 2: number analyzed (Participants) | 239 | 463 | 198 | 382
  MenY Before Vacc 2 | 100.0 [98.5 to 100.0] | 97.2 [95.2 to 98.5] | 100.0 [98.2 to 100.0] | 99.5 [98.1 to 99.9]

66. Secondary Outcome: Stage1: Percentage of Participants With hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY Titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, and >=1:128 for ACWY Test Strains Before Vaccination 1 and Before Vaccination 2: Groups 1, 2, 3 and 4
Description: Percentage of participants who achieved an hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY titer >=1:4, >= :8, >=1:16, >=1:32, >=1:64, >=1:128 for ACWY test strains was reported in this outcome measure.
Time Frame: Before Vaccination 1 (Vacc 1) [Day 1], Before Vaccination 2 (Vacc 2) [173 to 194 Days After Visit 1]
Population: as for outcome 56
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 272 | 534 | 271 | 523
Percentage of participants
  MenA Before Vacc 1 >=1:4: number analyzed (Participants) | 270 | 528 | 219 | 418
  MenA Before Vacc 1 >=1:4 | 26.3 [21.1 to 32.0] | 33.3 [29.3 to 37.5] | 64.4 [57.7 to 70.7] | 65.8 [61.0 to 70.3]
  MenA Before Vacc 1 >=1:8: number analyzed (Participants) | 270 | 528 | 219 | 418
  MenA Before Vacc 1 >=1:8 | 15.9 [11.8 to 20.8] | 22.9 [19.4 to 26.7] | 53.9 [47.0 to 60.6] | 52.6 [47.7 to 57.5]
  MenA Before Vacc 1 >=1:16: number analyzed (Participants) | 270 | 528 | 219 | 418
  MenA Before Vacc 1 >=1:16 | 14.4 [10.5 to 19.2] | 18.0 [14.8 to 21.5] | 40.2 [33.6 to 47.0] | 41.6 [36.9 to 46.5]
  MenA Before Vacc 1 >=1:32: number analyzed (Participants) | 270 | 528 | 219 | 418
  MenA Before Vacc 1 >=1:32 | 8.5 [5.5 to 12.5] | 10.6 [8.1 to 13.6] | 24.2 [18.7 to 30.4] | 22.0 [18.1 to 26.3]
  MenA Before Vacc 1 >=1:64: number analyzed (Participants) | 270 | 528 | 219 | 418
  MenA Before Vacc 1 >=1:64 | 5.2 [2.9 to 8.5] | 5.5 [3.7 to 7.8] | 12.8 [8.7 to 17.9] | 15.1 [11.8 to 18.9]
  MenA Before Vacc 1 >=1:128: number analyzed (Participants) | 270 | 528 | 219 | 418
  MenA Before Vacc 1 >=1:128 | 3.0 [1.3 to 5.8] | 4.0 [2.5 to 6.0] | 7.8 [4.6 to 12.1] | 6.2 [4.1 to 9.0]
  MenA Before Vacc 2 >=1:4: number analyzed (Participants) | 238 | 463 | 200 | 385
  MenA Before Vacc 2 >=1:4 | 93.3 [89.3 to 96.1] | 88.3 [85.1 to 91.1] | 99.0 [96.4 to 99.9] | 98.4 [96.6 to 99.4]
  MenA Before Vacc 2 >=1:8: number analyzed (Participants) | 238 | 463 | 200 | 385
  MenA Before Vacc 2 >=1:8 | 91.6 [87.3 to 94.8] | 86.2 [82.7 to 89.2] | 99.0 [96.4 to 99.9] | 98.4 [96.6 to 99.4]
  MenA Before Vacc 2 >=1:16: number analyzed (Participants) | 238 | 463 | 200 | 385
  MenA Before Vacc 2 >=1:16 | 87.4 [82.5 to 91.3] | 81.9 [78.0 to 85.3] | 98.0 [95.0 to 99.5] | 98.4 [96.6 to 99.4]
  MenA Before Vacc 2 >=1:32: number analyzed (Participants) | 238 | 463 | 200 | 385
  MenA Before Vacc 2 >=1:32 | 72.3 [66.1 to 77.9] | 66.3 [61.8 to 70.6] | 95.5 [91.6 to 97.9] | 96.1 [93.7 to 97.8]
  MenA Before Vacc 2 >=1:64: number analyzed (Participants) | 238 | 463 | 200 | 385
  MenA Before Vacc 2 >=1:64 | 44.5 [38.1 to 51.1] | 50.5 [45.9 to 55.2] | 85.0 [79.3 to 89.6] | 88.8 [85.3 to 91.8]
  MenA Before Vacc 2 >=1:128: number analyzed (Participants) | 238 | 463 | 200 | 385
  MenA Before Vacc 2 >=1:128 | 25.2 [19.8 to 31.2] | 33.5 [29.2 to 38.0] | 64.0 [56.9 to 70.6] | 75.3 [70.7 to 79.6]
  MenC Before Vacc 1 >=1:4: number analyzed (Participants) | 267 | 526 | 264 | 511
  MenC Before Vacc 1 >=1:4 | 63.7 [57.6 to 69.4] | 59.7 [55.4 to 63.9] | 76.1 [70.5 to 81.1] | 78.3 [74.4 to 81.8]
  MenC Before Vacc 1 >=1:8: number analyzed (Participants) | 267 | 526 | 264 | 511
  MenC Before Vacc 1 >=1:8 | 38.6 [32.7 to 44.7] | 39.0 [34.8 to 43.3] | 59.5 [53.3 to 65.4] | 61.1 [56.7 to 65.3]
  MenC Before Vacc 1 >=1:16: number analyzed (Participants) | 267 | 526 | 264 | 511
  MenC Before Vacc 1 >=1:16 | 24.3 [19.3 to 29.9] | 24.5 [20.9 to 28.4] | 42.0 [36.0 to 48.3] | 44.4 [40.1 to 48.9]
  MenC Before Vacc 1 >=1:32: number analyzed (Participants) | 267 | 526 | 264 | 511
  MenC Before Vacc 1 >=1:32 | 12.0 [8.3 to 16.5] | 12.5 [9.8 to 15.7] | 26.9 [21.6 to 32.7] | 29.7 [25.8 to 33.9]
  MenC Before Vacc 1 >=1:64: number analyzed (Participants) | 267 | 526 | 264 | 511
  MenC Before Vacc 1 >=1:64 | 5.2 [2.9 to 8.6] | 6.8 [4.8 to 9.3] | 15.9 [11.7 to 20.9] | 18.2 [14.9 to 21.8]
  MenC Before Vacc 1 >=1:128: number analyzed (Participants) | 267 | 526 | 264 | 511
  MenC Before Vacc 1 >=1:128 | 4.5 [2.3 to 7.7] | 4.0 [2.5 to 6.0] | 6.8 [4.1 to 10.6] | 9.2 [6.8 to 12.0]
  MenC Before Vacc 2 >=1:4: number analyzed (Participants) | 239 | 460 | 243 | 474
  MenC Before Vacc 2 >=1:4 | 95.0 [91.4 to 97.4] | 85.9 [82.3 to 88.9] | 99.6 [97.7 to 100.0] | 99.4 [98.2 to 99.9]
  MenC Before Vacc 2 >=1:8: number analyzed (Participants) | 239 | 460 | 243 | 474
  MenC Before Vacc 2 >=1:8 | 92.9 [88.9 to 95.8] | 76.5 [72.4 to 80.3] | 98.4 [95.8 to 99.5] | 98.3 [96.7 to 99.3]
  MenC Before Vacc 2 >=1:16: number analyzed (Participants) | 239 | 460 | 243 | 474
  MenC Before Vacc 2 >=1:16 | 84.9 [79.8 to 89.2] | 68.3 [63.8 to 72.5] | 98.4 [95.8 to 99.5] | 97.3 [95.4 to 98.5]
  MenC Before Vacc 2 >=1:32: number analyzed (Participants) | 239 | 460 | 243 | 474
  MenC Before Vacc 2 >=1:32 | 68.2 [61.9 to 74.1] | 52.4 [47.7 to 57.0] | 95.9 [92.6 to 98.0] | 91.6 [88.7 to 93.9]
  MenC Before Vacc 2 >=1:64: number analyzed (Participants) | 239 | 460 | 243 | 474
  MenC Before Vacc 2 >=1:64 | 53.1 [46.6 to 59.6] | 39.3 [34.9 to 44.0] | 92.6 [88.5 to 95.6] | 81.2 [77.4 to 84.6]
  MenC Before Vacc 2 >=1:128: number analyzed (Participants) | 239 | 460 | 243 | 474
  MenC Before Vacc 2 >=1:128 | 36.8 [30.7 to 43.3] | 27.8 [23.8 to 32.2] | 78.2 [72.5 to 83.2] | 66.2 [61.8 to 70.5]
  MenW Before Vacc 1 >=1:4: number analyzed (Participants) | 268 | 527 | 218 | 418
  MenW Before Vacc 1 >=1:4 | 47.8 [41.6 to 53.9] | 50.5 [46.1 to 54.8] | 83.0 [77.4 to 87.8] | 76.3 [71.9 to 80.3]
  MenW Before Vacc 1 >=1:8: number analyzed (Participants) | 268 | 527 | 218 | 418
  MenW Before Vacc 1 >=1:8 | 32.1 [26.5 to 38.0] | 34.5 [30.5 to 38.8] | 61.9 [55.1 to 68.4] | 60.8 [55.9 to 65.5]
  MenW Before Vacc 1 >=1:16: number analyzed (Participants) | 268 | 527 | 218 | 418
  MenW Before Vacc 1 >=1:16 | 23.9 [18.9 to 29.4] | 22.8 [19.3 to 26.6] | 37.6 [31.2 to 44.4] | 39.7 [35.0 to 44.6]
  MenW Before Vacc 1 >=1:32: number analyzed (Participants) | 268 | 527 | 218 | 418
  MenW Before Vacc 1 >=1:32 | 10.8 [7.4 to 15.2] | 13.7 [10.8 to 16.9] | 20.2 [15.1 to 26.1] | 21.8 [17.9 to 26.0]
  MenW Before Vacc 1 >=1:64: number analyzed (Participants) | 268 | 527 | 218 | 418
  MenW Before Vacc 1 >=1:64 | 7.5 [4.6 to 11.3] | 6.3 [4.3 to 8.7] | 9.2 [5.7 to 13.8] | 11.2 [8.4 to 14.7]
  MenW Before Vacc 1 >=1:128: number analyzed (Participants) | 268 | 527 | 218 | 418
  MenW Before Vacc 1 >=1:128 | 4.5 [2.3 to 7.7] | 1.5 [0.7 to 3.0] | 5.5 [2.9 to 9.4] | 6.2 [4.1 to 9.0]
  MenW Before Vacc 2 >=1:4: number analyzed (Participants) | 242 | 467 | 199 | 385
  MenW Before Vacc 2 >=1:4 | 99.2 [97.0 to 99.9] | 96.6 [94.5 to 98.0] | 100.0 [98.2 to 100.0] | 99.0 [97.4 to 99.7]
  MenW Before Vacc 2 >=1:8: number analyzed (Participants) | 242 | 467 | 199 | 385
  MenW Before Vacc 2 >=1:8 | 99.2 [97.0 to 99.9] | 91.0 [88.0 to 93.4] | 100.0 [98.2 to 100.0] | 99.0 [97.4 to 99.7]
  MenW Before Vacc 2 >=1:16: number analyzed (Participants) | 242 | 467 | 199 | 385
  MenW Before Vacc 2 >=1:16 | 95.5 [92.0 to 97.7] | 82.7 [78.9 to 86.0] | 99.5 [97.2 to 100.0] | 97.7 [95.6 to 98.9]
  MenW Before Vacc 2 >=1:32: number analyzed (Participants) | 242 | 467 | 199 | 385
  MenW Before Vacc 2 >=1:32 | 78.5 [72.8 to 83.5] | 64.2 [59.7 to 68.6] | 98.5 [95.7 to 99.7] | 95.8 [93.3 to 97.6]
  MenW Before Vacc 2 >=1:64: number analyzed (Participants) | 242 | 467 | 199 | 385
  MenW Before Vacc 2 >=1:64 | 56.6 [50.1 to 62.9] | 41.1 [36.6 to 45.7] | 95.5 [91.6 to 97.9] | 89.1 [85.5 to 92.0]
  MenW Before Vacc 2 >=1:128: number analyzed (Participants) | 242 | 467 | 199 | 385
  MenW Before Vacc 2 >=1:128 | 34.3 [28.3 to 40.6] | 24.2 [20.4 to 28.3] | 84.4 [78.6 to 89.2] | 79.0 [74.5 to 82.9]
  MenY Before Vacc 1 >=1:4: number analyzed (Participants) | 265 | 528 | 219 | 421
  MenY Before Vacc 1 >=1:4 | 67.2 [61.2 to 72.8] | 70.3 [66.2 to 74.1] | 87.7 [82.6 to 91.7] | 89.5 [86.2 to 92.3]
  MenY Before Vacc 1 >=1:8: number analyzed (Participants) | 265 | 528 | 219 | 421
  MenY Before Vacc 1 >=1:8 | 54.0 [47.8 to 60.1] | 58.1 [53.8 to 62.4] | 79.9 [74.0 to 85.0] | 77.9 [73.6 to 81.8]
  MenY Before Vacc 1 >=1:16: number analyzed (Participants) | 265 | 528 | 219 | 421
  MenY Before Vacc 1 >=1:16 | 44.2 [38.1 to 50.4] | 46.6 [42.3 to 50.9] | 67.1 [60.5 to 73.3] | 65.8 [61.0 to 70.3]
  MenY Before Vacc 1 >=1:32: number analyzed (Participants) | 265 | 528 | 219 | 421
  MenY Before Vacc 1 >=1:32 | 21.1 [16.4 to 26.5] | 26.7 [23.0 to 30.7] | 38.4 [31.9 to 45.1] | 40.9 [36.1 to 45.7]
  MenY Before Vacc 1 >=1:64: number analyzed (Participants) | 265 | 528 | 219 | 421
  MenY Before Vacc 1 >=1:64 | 10.9 [7.5 to 15.3] | 11.2 [8.6 to 14.2] | 21.9 [16.6 to 28.0] | 20.2 [16.5 to 24.3]
  MenY Before Vacc 1 >=1:128: number analyzed (Participants) | 265 | 528 | 219 | 421
  MenY Before Vacc 1 >=1:128 | 4.9 [2.6 to 8.2] | 6.3 [4.3 to 8.7] | 10.0 [6.4 to 14.8] | 10.5 [7.7 to 13.8]
  MenY Before Vacc 2 >=1:4: number analyzed (Participants) | 239 | 463 | 198 | 382
  MenY Before Vacc 2 >=1:4 | 100.0 [98.5 to 100.0] | 98.9 [97.5 to 99.6] | 100.0 [98.2 to 100.0] | 99.5 [98.1 to 99.9]
  MenY Before Vacc 2 >=1:8: number analyzed (Participants) | 239 | 463 | 198 | 382
  MenY Before Vacc 2 >=1:8 | 100.0 [98.5 to 100.0] | 97.2 [95.2 to 98.5] | 100.0 [98.2 to 100.0] | 99.5 [98.1 to 99.9]
  MenY Before Vacc 2 >=1:16: number analyzed (Participants) | 239 | 463 | 198 | 382
  MenY Before Vacc 2 >=1:16 | 98.3 [95.8 to 99.5] | 92.9 [90.1 to 95.0] | 100.0 [98.2 to 100.0] | 99.2 [97.7 to 99.8]
  MenY Before Vacc 2 >=1:32: number analyzed (Participants) | 239 | 463 | 198 | 382
  MenY Before Vacc 2 >=1:32 | 87.0 [82.1 to 91.0] | 77.1 [73.0 to 80.9] | 99.0 [96.4 to 99.9] | 95.8 [93.3 to 97.6]
  MenY Before Vacc 2 >=1:64: number analyzed (Participants) | 239 | 463 | 198 | 382
  MenY Before Vacc 2 >=1:64 | 69.9 [63.6 to 75.6] | 56.2 [51.5 to 60.7] | 94.9 [90.9 to 97.6] | 88.5 [84.8 to 91.5]
  MenY Before Vacc 2 >=1:128: number analyzed (Participants) | 239 | 463 | 198 | 382
  MenY Before Vacc 2 >=1:128 | 41.0 [34.7 to 47.5] | 31.1 [26.9 to 35.5] | 86.4 [80.8 to 90.8] | 80.6 [76.3 to 84.5]

67. Secondary Outcome: Stage1: hSBA GMTs for ACWY Test Strains Before Vaccination 1 and Before Vaccination 2: Groups 1, 2, 3 and 4
Description: GMTs were calculated using all participants with valid and determinate hSBA titers at the given time point. LLOQ = 1:8 for all MenA, MenC, MenW, and MenY strains. Titers below the LLOQ were set to 0.5*LLOQ for analysis. Confidence intervals were back transformations of confidence levels based on the Student t distribution for the mean logarithm of the concentrations, or the mean of the ratio.
Time Frame: Before Vaccination 1 (Vacc 1) [Day 1], Before Vaccination 2 (Vacc 2) [173 to 194 Days After Visit 1]
Population: as for outcome 56
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 272 | 534 | 271 | 523
Titers
  MenA Before Vacc 1: number analyzed (Participants) | 270 | 528 | 219 | 418
  MenA Before Vacc 1 | 5.7 [5.1 to 6.3] | 6.3 [5.7 to 6.8] | 11.0 [9.3 to 13.0] | 10.7 [9.6 to 12.0]
  MenA Before Vacc 2: number analyzed (Participants) | 238 | 463 | 200 | 385
  MenA Before Vacc 2 | 42.7 [36.1 to 50.4] | 47.2 [40.8 to 54.5] | 158.7 [132.6 to 189.8] | 214.6 [187.7 to 245.3]
  MenC Before Vacc 1: number analyzed (Participants) | 267 | 526 | 264 | 511
  MenC Before Vacc 1 | 7.5 [6.6 to 8.5] | 7.5 [6.8 to 8.2] | 11.9 [10.2 to 13.8] | 13.4 [11.9 to 15.1]
  MenC Before Vacc 2: number analyzed (Participants) | 239 | 460 | 243 | 474
  MenC Before Vacc 2 | 61.5 [49.5 to 76.3] | 32.7 [27.8 to 38.5] | 253.1 [213.0 to 300.8] | 186.7 [161.9 to 215.2]
  MenW Before Vacc 1: number analyzed (Participants) | 268 | 527 | 218 | 418
  MenW Before Vacc 1 | 7.0 [6.2 to 7.9] | 7.0 [6.4 to 7.5] | 10.5 [9.1 to 12.2] | 11.0 [9.8 to 12.3]
  MenW Before Vacc 2: number analyzed (Participants) | 242 | 467 | 199 | 385
  MenW Before Vacc 2 | 62.6 [53.5 to 73.1] | 39.1 [34.4 to 44.5] | 376.8 [311.4 to 456.0] | 255.5 [221.4 to 295.0]
  MenY Before Vacc 1: number analyzed (Participants) | 265 | 528 | 219 | 421
  MenY Before Vacc 1 | 10.5 [9.1 to 12.1] | 11.5 [10.4 to 12.7] | 19.2 [16.3 to 22.5] | 19.0 [16.8 to 21.4]
  MenY Before Vacc 2: number analyzed (Participants) | 239 | 463 | 198 | 382
  MenY Before Vacc 2 | 83.6 [71.4 to 97.8] | 58.6 [52.0 to 66.0] | 395.2 [327.8 to 476.3] | 264.0 [228.5 to 305.0]

68. Secondary Outcome: Stage1: Percentage of Participants With hSBA Titer Level >=LLOQ for 4 Primary MenB Test Strains Before Vaccination 1 and Before Vaccination 2 (Group 1 and 3 Combined; Group 2 and 4 Combined)
Description: as for outcome 61
Time Frame: Before Vaccination 1 (Vacc 1) [Day 1], Before Vaccination 2 (Vacc 2) [173 to 194 Days After Visit 1]
Population: as for outcome 61
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Group 1+3 Combined (MenABCWY + Saline): Stage 1: ACWY-naive and experienced participants who received an intramuscular injection of 0.5 milliliter (mL) of Neisseria meningitidis groups A, B, C, W, and Y vaccine (MenABCWY) and 0.5 mL of saline at Month 0, participants received 0.5 mL of MenABCWY vaccine intramuscularly at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received 0.5 mL of MenABCWY vaccine (booster vaccination) intramuscularly at Month 54.
Arm/Group | Group 1+3 Combined (MenABCWY + Saline) | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 438 | 864
Percentage of participants
  PMB80 (A22) Before Vacc 1: number analyzed (Participants) | 427 | 839
  PMB80 (A22) Before Vacc 1 | 25.3 [21.2 to 29.7] | 25.1 [22.2 to 28.2]
  PMB80 (A22) Before Vacc 2: number analyzed (Participants) | 425 | 842
  PMB80 (A22) Before Vacc 2 | 41.6 [36.9 to 46.5] | 41.9 [38.6 to 45.3]
  PMB2001 (A56) Before Vacc 1: number analyzed (Participants) | 421 | 833
  PMB2001 (A56) Before Vacc 1 | 13.8 [10.6 to 17.4] | 12.8 [10.6 to 15.3]
  PMB2001 (A56) Before Vacc 2: number analyzed (Participants) | 412 | 811
  PMB2001 (A56) Before Vacc 2 | 52.2 [47.2 to 57.1] | 45.7 [42.3 to 49.2]
  PMB2948 (B24) Before Vacc 1: number analyzed (Participants) | 434 | 855
  PMB2948 (B24) Before Vacc 1 | 10.4 [7.7 to 13.6] | 11.9 [9.8 to 14.3]
  PMB2948 (B24) Before Vacc 2: number analyzed (Participants) | 430 | 843
  PMB2948 (B24) Before Vacc 2 | 26.5 [22.4 to 31.0] | 24.2 [21.3 to 27.2]
  PMB2707 (B44) Before Vacc 1: number analyzed (Participants) | 434 | 861
  PMB2707 (B44) Before Vacc 1 | 3.7 [2.1 to 5.9] | 4.5 [3.2 to 6.1]
  PMB2707 (B44) Before Vacc 2: number analyzed (Participants) | 421 | 843
  PMB2707 (B44) Before Vacc 2 | 18.8 [15.1 to 22.8] | 16.5 [14.0 to 19.2]

69. Secondary Outcome: Stage1: Percentage of Participants With hSBA Titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, and >=1:128 for Each of the 4 Primary MenB Test Strains Before Vaccination 1 and Before Vaccination 2 (Group 1 and 3 Combined; Group 2 and 4 Combined)
Description: Percentage of participants who achieved an hSBA titer >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, and >=1:128 for each of the 4 primary MenB test strains was reported in this outcome measure.
Time Frame: Before Vaccination 1 (Vacc 1) [Day 1], Before Vaccination 2 (Vacc 2) [173 to 194 Days After Visit 1]
Population: Stage 1 EIP analyzed. Here, "Overall Number of Participants Analyzed" signifies number of participants measured and analyzed for this outcome measure. "Number Analyzed" signifies number of participants with valid and determinate hSBA results for each strain at given time point. Analysis was planned for combined Group 1 and 3 and combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1+3 Combined (MenABCWY + Saline) | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 438 | 864
Percentage of participants
  PMB80 (A22) Before Vacc 1 >=1:4: number analyzed (Participants) | 427 | 839
  PMB80 (A22) Before Vacc 1 >=1:4 | 34.7 [30.1 to 39.4] | 36.6 [33.3 to 40.0]
  PMB80 (A22) Before Vacc 1 >=1:8: number analyzed (Participants) | 427 | 839
  PMB80 (A22) Before Vacc 1 >=1:8 | 31.9 [27.5 to 36.5] | 31.8 [28.7 to 35.1]
  PMB80 (A22) Before Vacc 1 >=1:16: number analyzed (Participants) | 427 | 839
  PMB80 (A22) Before Vacc 1 >=1:16 | 25.3 [21.2 to 29.7] | 25.1 [22.2 to 28.2]
  PMB80 (A22) Before Vacc 1 >=1:32: number analyzed (Participants) | 427 | 839
  PMB80 (A22) Before Vacc 1 >=1:32 | 11.0 [8.2 to 14.4] | 11.4 [9.4 to 13.8]
  PMB80 (A22) Before Vacc 1 >=1:64: number analyzed (Participants) | 427 | 839
  PMB80 (A22) Before Vacc 1 >=1:64 | 4.7 [2.9 to 7.1] | 4.4 [3.1 to 6.0]
  PMB80 (A22) Before Vacc 1 >=1:128: number analyzed (Participants) | 427 | 839
  PMB80 (A22) Before Vacc 1 >=1:128 | 1.4 [0.5 to 3.0] | 0.8 [0.3 to 1.7]
  PMB80 (A22) Before Vacc 2 >=1:4: number analyzed (Participants) | 425 | 842
  PMB80 (A22) Before Vacc 2 >=1:4 | 48.2 [43.4 to 53.1] | 49.8 [46.3 to 53.2]
  PMB80 (A22) Before Vacc 2 >=1:8: number analyzed (Participants) | 425 | 842
  PMB80 (A22) Before Vacc 2 >=1:8 | 44.5 [39.7 to 49.3] | 46.6 [43.1 to 50.0]
  PMB80 (A22) Before Vacc 2 >=1:16: number analyzed (Participants) | 425 | 842
  PMB80 (A22) Before Vacc 2 >=1:16 | 41.6 [36.9 to 46.5] | 41.9 [38.6 to 45.3]
  PMB80 (A22) Before Vacc 2 >=1:32: number analyzed (Participants) | 425 | 842
  PMB80 (A22) Before Vacc 2 >=1:32 | 23.5 [19.6 to 27.9] | 23.5 [20.7 to 26.5]
  PMB80 (A22) Before Vacc 2 >=1:64: number analyzed (Participants) | 425 | 842
  PMB80 (A22) Before Vacc 2 >=1:64 | 9.9 [7.2 to 13.1] | 9.0 [7.2 to 11.2]
  PMB80 (A22) Before Vacc 2 >=1:128: number analyzed (Participants) | 425 | 842
  PMB80 (A22) Before Vacc 2 >=1:128 | 2.6 [1.3 to 4.6] | 3.2 [2.1 to 4.6]
  PMB2001 (A56) Before Vacc 1 >=1:4: number analyzed (Participants) | 421 | 833
  PMB2001 (A56) Before Vacc 1 >=1:4 | 19.5 [15.8 to 23.6] | 17.5 [15.0 to 20.3]
  PMB2001 (A56) Before Vacc 1 >=1:8: number analyzed (Participants) | 421 | 833
  PMB2001 (A56) Before Vacc 1 >=1:8 | 13.8 [10.6 to 17.4] | 12.8 [10.6 to 15.3]
  PMB2001 (A56) Before Vacc 1 >=1:16: number analyzed (Participants) | 421 | 833
  PMB2001 (A56) Before Vacc 1 >=1:16 | 10.7 [7.9 to 14.0] | 11.0 [9.0 to 13.4]
  PMB2001 (A56) Before Vacc 1 >=1:32: number analyzed (Participants) | 421 | 833
  PMB2001 (A56) Before Vacc 1 >=1:32 | 6.7 [4.5 to 9.5] | 7.6 [5.9 to 9.6]
  PMB2001 (A56) Before Vacc 1 >=1:64: number analyzed (Participants) | 421 | 833
  PMB2001 (A56) Before Vacc 1 >=1:64 | 3.8 [2.2 to 6.1] | 4.3 [3.0 to 5.9]
  PMB2001 (A56) Before Vacc 1 >=1:128: number analyzed (Participants) | 421 | 833
  PMB2001 (A56) Before Vacc 1 >=1:128 | 2.9 [1.5 to 4.9] | 2.4 [1.5 to 3.7]
  PMB2001 (A56) Before Vacc 2 >=1:4: number analyzed (Participants) | 412 | 811
  PMB2001 (A56) Before Vacc 2 >=1:4 | 56.6 [51.6 to 61.4] | 50.6 [47.1 to 54.1]
  PMB2001 (A56) Before Vacc 2 >=1:8: number analyzed (Participants) | 412 | 811
  PMB2001 (A56) Before Vacc 2 >=1:8 | 52.2 [47.2 to 57.1] | 45.7 [42.3 to 49.2]
  PMB2001 (A56) Before Vacc 2 >=1:16: number analyzed (Participants) | 412 | 811
  PMB2001 (A56) Before Vacc 2 >=1:16 | 47.1 [42.2 to 52.0] | 41.2 [37.8 to 44.7]
  PMB2001 (A56) Before Vacc 2 >=1:32: number analyzed (Participants) | 412 | 811
  PMB2001 (A56) Before Vacc 2 >=1:32 | 35.2 [30.6 to 40.0] | 30.9 [27.8 to 34.3]
  PMB2001 (A56) Before Vacc 2 >=1:64: number analyzed (Participants) | 412 | 811
  PMB2001 (A56) Before Vacc 2 >=1:64 | 21.4 [17.5 to 25.6] | 19.0 [16.3 to 21.9]
  PMB2001 (A56) Before Vacc 2 >=1:128: number analyzed (Participants) | 412 | 811
  PMB2001 (A56) Before Vacc 2 >=1:128 | 10.0 [7.2 to 13.3] | 9.5 [7.6 to 11.7]
  PMB2948 (B24) Before Vacc 1 >=1:4: number analyzed (Participants) | 434 | 855
  PMB2948 (B24) Before Vacc 1 >=1:4 | 14.1 [10.9 to 17.7] | 14.6 [12.3 to 17.2]
  PMB2948 (B24) Before Vacc 1 >=1:8: number analyzed (Participants) | 434 | 855
  PMB2948 (B24) Before Vacc 1 >=1:8 | 10.4 [7.7 to 13.6] | 11.9 [9.8 to 14.3]
  PMB2948 (B24) Before Vacc 1 >=1:16: number analyzed (Participants) | 434 | 855
  PMB2948 (B24) Before Vacc 1 >=1:16 | 6.2 [4.1 to 8.9] | 8.2 [6.4 to 10.2]
  PMB2948 (B24) Before Vacc 1 >=1:32: number analyzed (Participants) | 434 | 855
  PMB2948 (B24) Before Vacc 1 >=1:32 | 3.7 [2.1 to 5.9] | 4.2 [3.0 to 5.8]
  PMB2948 (B24) Before Vacc 1 >=1:64: number analyzed (Participants) | 434 | 855
  PMB2948 (B24) Before Vacc 1 >=1:64 | 0.9 [0.3 to 2.3] | 2.3 [1.4 to 3.6]
  PMB2948 (B24) Before Vacc 1 >=1:128: number analyzed (Participants) | 434 | 855
  PMB2948 (B24) Before Vacc 1 >=1:128 | 0.2 [0.0 to 1.3] | 1.1 [0.5 to 2.0]
  PMB2948 (B24) Before Vacc 2 >=1:4: number analyzed (Participants) | 430 | 843
  PMB2948 (B24) Before Vacc 2 >=1:4 | 30.5 [26.1 to 35.1] | 28.0 [25.0 to 31.2]
  PMB2948 (B24) Before Vacc 2 >=1:8: number analyzed (Participants) | 430 | 843
  PMB2948 (B24) Before Vacc 2 >=1:8 | 26.5 [22.4 to 31.0] | 24.2 [21.3 to 27.2]
  PMB2948 (B24) Before Vacc 2 >=1:16: number analyzed (Participants) | 430 | 843
  PMB2948 (B24) Before Vacc 2 >=1:16 | 21.4 [17.6 to 25.6] | 20.2 [17.5 to 23.0]
  PMB2948 (B24) Before Vacc 2 >=1:32: number analyzed (Participants) | 430 | 843
  PMB2948 (B24) Before Vacc 2 >=1:32 | 11.2 [8.3 to 14.5] | 11.0 [9.0 to 13.3]
  PMB2948 (B24) Before Vacc 2 >=1:64: number analyzed (Participants) | 430 | 843
  PMB2948 (B24) Before Vacc 2 >=1:64 | 5.1 [3.2 to 7.6] | 5.7 [4.2 to 7.5]
  PMB2948 (B24) Before Vacc 2 >=1:128: number analyzed (Participants) | 430 | 843
  PMB2948 (B24) Before Vacc 2 >=1:128 | 2.3 [1.1 to 4.2] | 2.3 [1.4 to 3.5]
  PMB2707 (B44) Before Vacc 1 >=1:4: number analyzed (Participants) | 434 | 861
  PMB2707 (B44) Before Vacc 1 >=1:4 | 7.1 [4.9 to 10.0] | 7.2 [5.6 to 9.1]
  PMB2707 (B44) Before Vacc 1 >=1:8: number analyzed (Participants) | 434 | 861
  PMB2707 (B44) Before Vacc 1 >=1:8 | 3.7 [2.1 to 5.9] | 4.5 [3.2 to 6.1]
  PMB2707 (B44) Before Vacc 1 >=1:16: number analyzed (Participants) | 434 | 861
  PMB2707 (B44) Before Vacc 1 >=1:16 | 2.1 [1.0 to 3.9] | 3.3 [2.2 to 4.7]
  PMB2707 (B44) Before Vacc 1 >=1:32: number analyzed (Participants) | 434 | 861
  PMB2707 (B44) Before Vacc 1 >=1:32 | 0.9 [0.3 to 2.3] | 2.1 [1.2 to 3.3]
  PMB2707 (B44) Before Vacc 1 >=1:64: number analyzed (Participants) | 434 | 861
  PMB2707 (B44) Before Vacc 1 >=1:64 | 0.7 [0.1 to 2.0] | 1.2 [0.6 to 2.1]
  PMB2707 (B44) Before Vacc 1 >=1:128: number analyzed (Participants) | 434 | 861
  PMB2707 (B44) Before Vacc 1 >=1:128 | 0.5 [0.1 to 1.7] | 0.3 [0.1 to 1.0]
  PMB2707 (B44) Before Vacc 2 >=1:4: number analyzed (Participants) | 421 | 843
  PMB2707 (B44) Before Vacc 2 >=1:4 | 29.2 [24.9 to 33.8] | 25.7 [22.8 to 28.8]
  PMB2707 (B44) Before Vacc 2 >=1:8: number analyzed (Participants) | 421 | 843
  PMB2707 (B44) Before Vacc 2 >=1:8 | 18.8 [15.1 to 22.8] | 16.5 [14.0 to 19.2]
  PMB2707 (B44) Before Vacc 2 >=1:16: number analyzed (Participants) | 421 | 843
  PMB2707 (B44) Before Vacc 2 >=1:16 | 13.5 [10.4 to 17.2] | 11.7 [9.6 to 14.1]
  PMB2707 (B44) Before Vacc 2 >=1:32: number analyzed (Participants) | 421 | 843
  PMB2707 (B44) Before Vacc 2 >=1:32 | 7.6 [5.3 to 10.6] | 5.8 [4.3 to 7.6]
  PMB2707 (B44) Before Vacc 2 >=1:64: number analyzed (Participants) | 421 | 843
  PMB2707 (B44) Before Vacc 2 >=1:64 | 3.3 [1.8 to 5.5] | 2.8 [1.8 to 4.2]
  PMB2707 (B44) Before Vacc 2 >=1:128: number analyzed (Participants) | 421 | 843
  PMB2707 (B44) Before Vacc 2 >=1:128 | 0.7 [0.1 to 2.1] | 1.4 [0.7 to 2.5]

70. Secondary Outcome: Stage1: hSBA GMTs for Each of the 4 Primary MenB Test Strains Before Vaccination 1 and Before Vaccination 2 (Group 1 and 3 Combined; Group 2 and 4 Combined)
Description: GMTs were calculated using all participants with valid and determinate hSBA titers at the given time point. LLOQ =1:16 for A22; 1:8 for A56, B24, and B44. Titers below the LLOQ were set to 0.5*LLOQ for analysis. CIs were back transformations of confidence levels based on the Student t distribution for the mean logarithm of the hSBA titers.
Time Frame: Before Vaccination 1 (Vacc 1) [Day 1], Before Vaccination 2 (Vacc 2) [173 to 194 Days After Visit 1]
Population: Stage 1 EIP analyzed. Here, "Overall Number of Participants Analyzed" signifies number of participants measured and analyzed for this outcome measure. "Number Analyzed" signifies number of participants with valid and determinate hSBA results for each of the 4 strains at given time point. Analysis was planned for combined Group 1 and 3 and combined Group 2 and 4.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1+3 Combined (MenABCWY + Saline) | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 438 | 864
Titers
  PMB80 (A22), Before vacc 1: number analyzed (Participants) | 427 | 839
  PMB80 (A22), Before vacc 1 | 10.8 [10.2 to 11.5] | 10.7 [10.3 to 11.1]
  PMB80 (A22), Before vacc 2: number analyzed (Participants) | 425 | 842
  PMB80 (A22), Before vacc 2 | 13.7 [12.8 to 14.8] | 13.8 [13.1 to 14.5]
  PMB2001 (A56), Before vacc 1: number analyzed (Participants) | 421 | 833
  PMB2001 (A56), Before vacc 1 | 5.2 [4.9 to 5.7] | 5.3 [5.0 to 5.6]
  PMB2001 (A56), Before vacc 2: number analyzed (Participants) | 412 | 811
  PMB2001 (A56), Before vacc 2 | 13.0 [11.4 to 14.8] | 11.4 [10.4 to 12.5]
  PMB2948 (B24), Before vacc 1: number analyzed (Participants) | 434 | 855
  PMB2948 (B24), Before vacc 1 | 4.6 [4.4 to 4.9] | 4.9 [4.7 to 5.1]
  PMB2948 (B24), Before vacc 2: number analyzed (Participants) | 430 | 843
  PMB2948 (B24), Before vacc 2 | 6.3 [5.8 to 6.9] | 6.2 [5.9 to 6.6]
  PMB2707 (B44), Before vacc 1: number analyzed (Participants) | 434 | 861
  PMB2707 (B44), Before vacc 1 | 4.2 [4.1 to 4.4] | 4.3 [4.2 to 4.5]
  PMB2707 (B44), Before vacc 2: number analyzed (Participants) | 421 | 843
  PMB2707 (B44), Before vacc 2 | 5.4 [5.1 to 5.8] | 5.3 [5.0 to 5.5]

71. Secondary Outcome: Stage2: Percentage of Participants With hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY Titers >=1:8 (or LLOQ if Higher) for ACWY Test Strains During Persistence Phase: Groups 1, 2, 3 and 4
Description: as for outcome 55
Time Frame: 12, 24, 36 and 48 months after Vaccination 2 (Vacc 2)
Population: Stage 2 mITT population included all participants who signed the ICD at Month 18 and who had at least 1 valid and determinate primary strain MenB or MenA/C/W/Y assay result available in Stage 2. "Overall Number of Participants Analyzed": participants who were measured and analyzed for the outcome measure and 'Number Analyzed' signifies number of participants with valid and determinate hSBA results for ACWY test strains at the given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced) | Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
Number analyzed (Participants) | 112 | 64 | 101 | 73
Percentage of participants
  MenA 12 Months after Vacc 2: number analyzed (Participants) | 112 | 59 | 48 | 22
  MenA 12 Months after Vacc 2 | 91.1 [84.2 to 95.6] | 71.2 [57.9 to 82.2] | 97.9 [88.9 to 99.9] | 100.0 [84.6 to 100.0]
  MenA 24 Months after Vacc 2: number analyzed (Participants) | 101 | 60 | 61 | 37
  MenA 24 Months after Vacc 2 | 88.1 [80.2 to 93.7] | 70.0 [56.8 to 81.2] | 100.0 [94.1 to 100.0] | 100.0 [90.5 to 100.0]
  MenA 36 Months after Vacc 2: number analyzed (Participants) | 95 | 54 | 57 | 33
  MenA 36 Months after Vacc 2 | 88.4 [80.2 to 94.1] | 72.2 [58.4 to 83.5] | 100.0 [93.7 to 100.0] | 97.0 [84.2 to 99.9]
  MenA 48 Months after Vacc 2: number analyzed (Participants) | 71 | 41 | 40 | 23
  MenA 48 Months after Vacc 2 | 81.7 [70.7 to 89.9] | 63.4 [46.9 to 77.9] | 100.0 [91.2 to 100.0] | 100.0 [85.2 to 100.0]
  MenC 12 Months after Vacc 2: number analyzed (Participants) | 112 | 62 | 54 | 23
  MenC 12 Months after Vacc 2 | 76.8 [67.9 to 84.2] | 51.6 [38.6 to 64.5] | 96.3 [87.3 to 99.5] | 91.3 [72.0 to 98.9]
  MenC 24 Months after Vacc 2: number analyzed (Participants) | 101 | 61 | 97 | 71
  MenC 24 Months after Vacc 2 | 75.2 [65.7 to 83.3] | 47.5 [34.6 to 60.7] | 96.9 [91.2 to 99.4] | 94.4 [86.2 to 98.4]
  MenC 36 Months after Vacc 2: number analyzed (Participants) | 95 | 54 | 96 | 67
  MenC 36 Months after Vacc 2 | 67.4 [57.0 to 76.6] | 44.4 [30.9 to 58.6] | 96.9 [91.1 to 99.4] | 95.5 [87.5 to 99.1]
  MenC 48 Months after Vacc 2: number analyzed (Participants) | 71 | 42 | 76 | 58
  MenC 48 Months after Vacc 2 | 62.0 [49.7 to 73.2] | 38.1 [23.6 to 54.4] | 98.7 [92.9 to 100.0] | 89.7 [78.8 to 96.1]
  MenW 12 Months after Vacc 2: number analyzed (Participants) | 112 | 62 | 48 | 22
  MenW 12 Months after Vacc 2 | 99.1 [95.1 to 100.0] | 83.9 [72.3 to 92.0] | 100.0 [92.6 to 100.0] | 95.5 [77.2 to 99.9]
  MenW 24 Months after Vacc 2: number analyzed (Participants) | 103 | 61 | 61 | 37
  MenW 24 Months after Vacc 2 | 99.0 [94.7 to 100.0] | 78.7 [66.3 to 88.1] | 100.0 [94.1 to 100.0] | 94.6 [81.8 to 99.3]
  MenW 36 Months after Vacc 2: number analyzed (Participants) | 97 | 54 | 57 | 33
  MenW 36 Months after Vacc 2 | 94.8 [88.4 to 98.3] | 77.8 [64.4 to 88.0] | 100.0 [93.7 to 100.0] | 97.0 [84.2 to 99.9]
  MenW 48 Months after Vacc 2: number analyzed (Participants) | 70 | 41 | 40 | 23
  MenW 48 Months after Vacc 2 | 91.4 [82.3 to 96.8] | 70.7 [54.5 to 83.9] | 100.0 [91.2 to 100.0] | 91.3 [72.0 to 98.9]
  MenY 12 Months after Vacc 2: number analyzed (Participants) | 112 | 62 | 48 | 22
  MenY 12 Months after Vacc 2 | 100.0 [96.8 to 100.0] | 98.4 [91.3 to 100.0] | 100.0 [92.6 to 100.0] | 100.0 [84.6 to 100.0]
  MenY 24 Months after Vacc 2: number analyzed (Participants) | 102 | 61 | 61 | 37
  MenY 24 Months after Vacc 2 | 100.0 [96.4 to 100.0] | 93.4 [84.1 to 98.2] | 100.0 [94.1 to 100.0] | 100.0 [90.5 to 100.0]
  MenY 36 Months after Vacc 2: number analyzed (Participants) | 97 | 54 | 57 | 33
  MenY 36 Months after Vacc 2 | 100.0 [96.3 to 100.0] | 90.7 [79.7 to 96.9] | 100.0 [93.7 to 100.0] | 100.0 [84.2 to 100.0]
  MenY 48 Months after Vacc 2: number analyzed (Participants) | 71 | 42 | 40 | 22
  MenY 48 Months after Vacc 2 | 100.0 [94.9 to 100.0] | 95.2 [83.8 to 99.4] | 100.0 [91.2 to 100.0] | 100.0 [84.6 to 100.0]

72. Secondary Outcome: Stage2: Percentage of Participants With hSBA Titer Level >=LLOQ for 4 Primary MenB Test Strains During Persistence Phase (Group 1 and 3 Combined; Group 2 and 4 Combined)
Description: as for outcome 61
Time Frame: 12, 24, 36 and 48 months after Vaccination 2 (Vacc 2)
Population: Stage 2 mITT population analyzed. "Overall Number of Participants Analyzed": participants who were measured and analyzed for the outcome measure and 'Number Analyzed' signifies number of participants with valid and determinate hSBA results on all 4 strains at the given time point. Analysis planned for combined Group 1 and 3, and Group 1 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1+3 Combined (MenABCWY + Saline) | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 213 | 137
Percentage of participants
  PMB80 (A22) 12 months after Vacc 2: number analyzed (Participants) | 162 | 83
  PMB80 (A22) 12 months after Vacc 2 | 32.7 [25.6 to 40.5] | 26.5 [17.4 to 37.3]
  PMB80 (A22) 24 months after Vacc 2: number analyzed (Participants) | 196 | 128
  PMB80 (A22) 24 months after Vacc 2 | 36.7 [30.0 to 43.9] | 28.9 [21.2 to 37.6]
  PMB80 (A22) 36 months after Vacc 2: number analyzed (Participants) | 185 | 116
  PMB80 (A22) 36 months after Vacc 2 | 29.2 [22.8 to 36.3] | 25.9 [18.2 to 34.8]
  PMB80 (A22) 48 months after Vacc 2: number analyzed (Participants) | 139 | 94
  PMB80 (A22) 48 months after Vacc 2 | 28.1 [20.8 to 36.3] | 31.9 [22.7 to 42.3]
  PMB2001 (A56) 12 months after Vacc 2: number analyzed (Participants) | 162 | 84
  PMB2001 (A56) 12 months after Vacc 2 | 33.3 [26.1 to 41.2] | 32.1 [22.4 to 43.2]
  PMB2001 (A56) 24 months after Vacc 2: number analyzed (Participants) | 196 | 131
  PMB2001 (A56) 24 months after Vacc 2 | 34.7 [28.1 to 41.8] | 33.6 [25.6 to 42.4]
  PMB2001 (A56) 36 months after Vacc 2: number analyzed (Participants) | 186 | 118
  PMB2001 (A56) 36 months after Vacc 2 | 29.0 [22.6 to 36.1] | 33.9 [25.4 to 43.2]
  PMB2001 (A56) 48 months after Vacc 2: number analyzed (Participants) | 145 | 98
  PMB2001 (A56) 48 months after Vacc 2 | 34.5 [26.8 to 42.8] | 29.6 [20.8 to 39.7]
  PMB2948 (B24) 12 months after Vacc 2: number analyzed (Participants) | 165 | 85
  PMB2948 (B24) 12 months after Vacc 2 | 30.9 [24.0 to 38.6] | 28.2 [19.0 to 39.0]
  PMB2948 (B24) 24 months after Vacc 2: number analyzed (Participants) | 196 | 131
  PMB2948 (B24) 24 months after Vacc 2 | 33.2 [26.6 to 40.2] | 27.5 [20.0 to 36.0]
  PMB2948 (B24) 36 months after Vacc 2: number analyzed (Participants) | 192 | 120
  PMB2948 (B24) 36 months after Vacc 2 | 35.4 [28.7 to 42.6] | 28.3 [20.5 to 37.3]
  PMB2948 (B24) 48 months after Vacc 2: number analyzed (Participants) | 145 | 98
  PMB2948 (B24) 48 months after Vacc 2 | 36.6 [28.7 to 44.9] | 26.5 [18.1 to 36.4]
  PMB2707 (B44) 12 months after Vacc 2: number analyzed (Participants) | 166 | 85
  PMB2707 (B44) 12 months after Vacc 2 | 18.7 [13.1 to 25.4] | 15.3 [8.4 to 24.7]
  PMB2707 (B44) 24 months after Vacc 2: number analyzed (Participants) | 200 | 132
  PMB2707 (B44) 24 months after Vacc 2 | 18.0 [12.9 to 24.0] | 18.2 [12.0 to 25.8]
  PMB2707 (B44) 36 months after Vacc 2: number analyzed (Participants) | 193 | 121
  PMB2707 (B44) 36 months after Vacc 2 | 20.2 [14.8 to 26.6] | 19.8 [13.1 to 28.1]
  PMB2707 (B44) 48 months after Vacc 2: number analyzed (Participants) | 148 | 99
  PMB2707 (B44) 48 months after Vacc 2 | 18.2 [12.4 to 25.4] | 16.2 [9.5 to 24.9]

73. Secondary Outcome: Stage2: Percentage of Participants With hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY Titers >=1:8 (or >=LLOQ if Higher) for ACWY Test Strains 1 Month After Booster Vaccination: Groups 1 and 3 (Separately)
Description: Percentage of participants who achieved an hSBA-MenA, hSBA-MenC, hSBA-MenW, and hSBA-MenY titer >=LLOQ for ACWY test strains (LLOQ = 1:8 for all MenA, MenC, MenW, and MenY strains) was reported in this outcome measure. Analysis was planned for Group 1 and 3 separately.
Time Frame: 1 month after booster vaccination
Population: Booster EIP=participants who were eligible(met Stage [S] 1 eligibility criteria, continually met S 2 eligibility criteria), received booster dose (BD) as intended (same vaccine as received in S 1), had blood drawn for assay testing in required time frame at Month 55, had valid and determinate (VAD) MenB or MenA/C/W/Y assay result after BD, no major protocol violations determined by medical monitor. 'Number Analyzed': participants with VAD hSBA results for ACWY test strains at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 60 | 70
Percentage of participants
  MenA: number analyzed (Participants) | 60 | 33
  MenA | 100.0 [94.0 to 100.0] | 100.0 [89.4 to 100.0]
  MenC | 100.0 [94.0 to 100.0] | 100.0 [94.9 to 100.0]
  MenW: number analyzed (Participants) | 60 | 33
  MenW | 100.0 [94.0 to 100.0] | 100.0 [89.4 to 100.0]
  MenY: number analyzed (Participants) | 60 | 33
  MenY | 100.0 [94.0 to 100.0] | 100.0 [89.4 to 100.0]

74. Secondary Outcome: Stage2: Percentage of Participants With hSBA Titer Level >=LLOQ for 4 Primary MenB Test Strains 1 Month After Booster Vaccination (Group 1 and 3 Combined; Group 2 and 4 Combined)
Description: as for outcome 61
Time Frame: 1 month after booster vaccination
Population: Booster EIP analyzed. Here, "Overall Number of Participants analyzed" signifies number of participants who were measured and analyzed for this outcome measure. 'Number Analyzed'=number of participants with VAD hSBA results for ACWY test strains at given time point. Analysis was planned for combined Group 1 and 3 and combined Group 2 and 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1+3 Combined (MenABCWY + Saline) | Groups 2+4 Combined (Bivalent rLP2086 + MenACWY-CRM)
Number analyzed (Participants) | 130 | 88
Percentage of participants
  PMB80 (A22): number analyzed (Participants) | 122 | 81
  PMB80 (A22) | 95.1 [89.6 to 98.2] | 93.8 [86.2 to 98.0]
  PMB2001 (A56): number analyzed (Participants) | 124 | 86
  PMB2001 (A56) | 100.0 [97.1 to 100.0] | 98.8 [93.7 to 100.0]
  PMB2948 (B24): number analyzed (Participants) | 123 | 84
  PMB2948 (B24) | 95.1 [89.7 to 98.2] | 95.2 [88.3 to 98.7]
  PMB2707 (B44): number analyzed (Participants) | 128 | 86
  PMB2707 (B44) | 99.2 [95.7 to 100.0] | 98.8 [93.7 to 100.0]

75. Secondary Outcome: Stage1: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1: Group 1 and Group 3
Description: as for outcome 3
Time Frame: 7 days after Vaccination 1 (Vacc 1)
Population: Vaccination 1 safety population included participants who received the first dose of investigational product (MenABCWY+saline or bivalent rLP2086+MenACWY-CRM) at Visit 1 (Month 0), and for whom safety information from Visit 1 (Month 0) to prior to Visit 3 (Month 6) was available. Here, 'Number of Participants Analyzed' signifies number of participants measured and analyzed for this outcome measure. Analysis was planned for Group 1 and 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 269 | 269
Percentage of participants
  Redness: Any | 19.7 [15.1 to 25.0] | 14.9 [10.8 to 19.7]
  Redness: Mild | 7.4 [4.6 to 11.2] | 5.6 [3.2 to 9.0]
  Redness: Moderate | 10.0 [6.7 to 14.3] | 7.4 [4.6 to 11.2]
  Redness: Severe | 2.2 [0.8 to 4.8] | 1.9 [0.6 to 4.3]
  Swelling: Any | 20.8 [16.1 to 26.2] | 17.5 [13.1 to 22.5]
  Swelling: Mild | 9.3 [6.1 to 13.4] | 8.6 [5.5 to 12.6]
  Swelling: Moderate | 10.4 [7.0 to 14.7] | 8.6 [5.5 to 12.6]
  Swelling: Severe | 1.1 [0.2 to 3.2] | 0.4 [0.0 to 2.1]
  Pain at injection site: Any | 89.2 [84.9 to 92.7] | 90.3 [86.2 to 93.6]
  Pain at injection site: Mild | 37.2 [31.4 to 43.3] | 45.4 [39.3 to 51.5]
  Pain at injection site: Moderate | 45.7 [39.7 to 51.9] | 40.1 [34.2 to 46.3]
  Pain at injection site: Severe: number analyzed (Participants) | 230 | 233
  Pain at injection site: Severe | 6.3 [3.7 to 9.9] | 4.8 [2.6 to 8.1]

76. Secondary Outcome: Stage1: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2: Group 1 and Group 3
Description: as for outcome 3
Time Frame: 7 days after Vaccination 2 (Vacc 2)
Population: Vaccination 2 safety population included participants who received the second dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 3 (Month 6), and for whom safety information from Visit 3 (Month 6) up to and including Visit 4 (month 7) was available. Here, 'Number of Participants Analyzed' signifies number of participants measured and analyzed for this outcome measure. Analysis was planned for Group 1 and 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 230 | 233
Percentage of participants
  Redness: Any | 23.0 [17.8 to 29.0] | 19.3 [14.4 to 25.0]
  Redness: Mild | 7.0 [4.0 to 11.1] | 6.9 [4.0 to 10.9]
  Redness: Moderate | 11.7 [7.9 to 16.6] | 9.0 [5.7 to 13.4]
  Redness: Severe | 4.3 [2.1 to 7.9] | 3.4 [1.5 to 6.7]
  Swelling: Any | 19.1 [14.3 to 24.8] | 18.0 [13.3 to 23.6]
  Swelling: Mild | 8.7 [5.4 to 13.1] | 5.6 [3.0 to 9.4]
  Swelling: Moderate | 10.0 [6.4 to 14.6] | 11.2 [7.4 to 15.9]
  Swelling: Severe | 0.4 [0.0 to 2.4] | 1.3 [0.3 to 3.7]
  Pain at injection site: Any | 85.2 [80.0 to 89.5] | 83.7 [78.3 to 88.2]
  Pain at injection site: Mild | 34.3 [28.2 to 40.9] | 37.8 [31.5 to 44.3]
  Pain at injection site: Moderate | 47.0 [40.4 to 53.6] | 38.2 [31.9 to 44.8]
  Pain at injection site: Severe | 3.9 [1.8 to 7.3] | 7.7 [4.6 to 11.9]

77. Secondary Outcome: Stage1: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1: Group 1 and Group 3
Description: Systemic events fever, vomiting, diarrhea, headache, fatigue, chills, muscle pain and joint pain were recorded in an e-diary. Fever was defined as >=38.0 degree C and categorized to 38.0 to 38.4 degree C, 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and >40.0 degree C. Headache, fatigue, chills, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily activity). Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required IV hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 in 24 hours).
Time Frame: 7 days after Vaccination 1 (Vacc 1)
Population: as for outcome 75
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 269 | 269
Percentage of participants
  Fever: >= 38.0 degree C | 7.4 [4.6 to 11.2] | 5.2 [2.9 to 8.6]
  Fever: 38.0 to 38.4 degree C | 4.1 [2.1 to 7.2] | 4.1 [2.1 to 7.2]
  Fever: 38.4 to 38.9 degree C | 2.2 [0.8 to 4.8] | 0.7 [0.1 to 2.7]
  Fever: 38.9 to 40.0 degree C | 1.1 [0.2 to 3.2] | 0.4 [0.0 to 2.1]
  Fever: > 40.0 degree C | 0.0 [0.0 to 1.4] | 0.0 [0.0 to 1.4]
  Fatigue: Any | 56.5 [50.4 to 62.5] | 49.1 [42.9 to 55.2]
  Fatigue: Mild | 26.8 [21.6 to 32.5] | 27.9 [22.6 to 33.6]
  Fatigue: Moderate | 25.3 [20.2 to 30.9] | 17.5 [13.1 to 22.5]
  Fatigue: Severe | 4.5 [2.3 to 7.7] | 3.7 [1.8 to 6.7]
  Headache: Any | 48.3 [42.2 to 54.5] | 45.0 [38.9 to 51.1]
  Headache: Mild | 27.1 [21.9 to 32.9] | 29.4 [24.0 to 35.2]
  Headache: Moderate | 19.3 [14.8 to 24.6] | 14.1 [10.2 to 18.9]
  Headache: Severe | 1.9 [0.6 to 4.3] | 1.5 [0.4 to 3.8]
  Chills: Any | 20.1 [15.5 to 25.4] | 14.9 [10.8 to 19.7]
  Chills: Mild | 14.5 [10.5 to 19.3] | 9.3 [6.1 to 13.4]
  Chills: Moderate | 4.5 [2.3 to 7.7] | 4.8 [2.6 to 8.1]
  Chills: Severe | 1.1 [0.2 to 3.2] | 0.7 [0.1 to 2.7]
  Vomiting: Any | 2.6 [1.1 to 5.3] | 1.9 [0.6 to 4.3]
  Vomiting: Mild | 2.2 [0.8 to 4.8] | 1.9 [0.6 to 4.3]
  Vomiting: Moderate | 0.4 [0.0 to 2.1] | 0.0 [0.0 to 1.4]
  Vomiting: severe | 0.0 [0.0 to 1.4] | 0.0 [0.0 to 1.4]
  Diarrhea: Any | 12.3 [8.6 to 16.8] | 15.2 [11.2 to 20.1]
  Diarrhea: Mild | 10.0 [6.7 to 14.3] | 10.8 [7.3 to 15.1]
  Diarrhea: Moderate | 2.2 [0.8 to 4.8] | 4.5 [2.3 to 7.7]
  Diarrhea: Severe | 0.0 [0.0 to 1.4] | 0.0 [0.0 to 1.4]
  Muscle pain: Any | 29.0 [23.6 to 34.8] | 22.7 [17.8 to 28.2]
  Muscle pain: Mild | 17.1 [12.8 to 22.1] | 14.5 [10.5 to 19.3]
  Muscle pain: Moderate | 10.4 [7.0 to 14.7] | 7.1 [4.3 to 10.8]
  Muscle pain: Severe | 1.5 [0.4 to 3.8] | 1.1 [0.2 to 3.2]
  Joint pain: Any | 20.8 [16.1 to 26.2] | 18.2 [13.8 to 23.4]
  Joint pain: Mild | 13.0 [9.2 to 17.6] | 10.8 [7.3 to 15.1]
  Joint pain: Moderate | 7.8 [4.9 to 11.7] | 6.7 [4.0 to 10.4]
  Joint pain: Severe | 0.0 [0.0 to 1.4] | 0.7 [0.1 to 2.7]

78. Secondary Outcome: Stage1: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2: Group 1 and Group 3
Description: as for outcome 77
Time Frame: 7 days after Vaccination 2 (Vacc 2)
Population: as for outcome 76
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 230 | 233
Percentage of participants
  Fever: >= 38.0 degree C | 3.5 [1.5 to 6.7] | 1.7 [0.5 to 4.3]
  Fever: 38.0 to 38.4°C | 2.2 [0.7 to 5.0] | 0.9 [0.1 to 3.1]
  Fever: 38.5 to 38.9°C | 1.3 [0.3 to 3.8] | 0.9 [0.1 to 3.1]
  Fever: 39.0 to 40.0°C | 0.0 [0.0 to 1.6] | 0.0 [0.0 to 1.6]
  Fever: > 40.0°C | 0.0 [0.0 to 1.6] | 0.0 [0.0 to 1.6]
  Fatigue: Any | 49.6 [42.9 to 56.2] | 47.6 [41.1 to 54.3]
  Fatigue: Mild | 20.9 [15.8 to 26.7] | 26.2 [20.7 to 32.3]
  Fatigue: Moderate | 26.1 [20.5 to 32.3] | 18.9 [14.1 to 24.5]
  Fatigue: Severe | 2.6 [1.0 to 5.6] | 2.6 [1.0 to 5.5]
  Headache: Any | 41.7 [35.3 to 48.4] | 43.8 [37.3 to 50.4]
  Headache: Mild | 22.6 [17.4 to 28.6] | 26.6 [21.1 to 32.8]
  Headache: Moderate | 17.8 [13.1 to 23.4] | 13.3 [9.2 to 18.4]
  Headache: Severe | 1.3 [0.3 to 3.8] | 3.9 [1.8 to 7.2]
  Chills: Any | 20.9 [15.8 to 26.7] | 19.3 [14.4 to 25.0]
  Chills: Mild | 16.1 [11.6 to 21.5] | 11.6 [7.8 to 16.4]
  Chills: Moderate | 3.9 [1.8 to 7.3] | 5.2 [2.7 to 8.8]
  Chills: Severe | 0.9 [0.1 to 3.1] | 2.6 [1.0 to 5.5]
  Vomiting: Any | 1.7 [0.5 to 4.4] | 3.9 [1.8 to 7.2]
  Vomiting: Mild | 1.7 [0.5 to 4.4] | 3.4 [1.5 to 6.7]
  Vomiting: Moderate | 0.0 [0.0 to 1.6] | 0.4 [0.0 to 2.4]
  Vomiting: Severe | 0.0 [0.0 to 1.6] | 0.0 [0.0 to 1.6]
  Diarrhea: Any | 13.5 [9.3 to 18.6] | 8.2 [5.0 to 12.4]
  Diarrhea: Mild | 9.6 [6.1 to 14.1] | 5.2 [2.7 to 8.8]
  Diarrhea: Moderate | 3.9 [1.8 to 7.3] | 2.6 [1.0 to 5.5]
  Diarrhea: Severe | 0.0 [0.0 to 1.6] | 0.4 [0.0 to 2.4]
  Muscle pain: Any | 24.8 [19.3 to 30.9] | 19.3 [14.4 to 25.0]
  Muscle pain: Mild | 13.0 [9.0 to 18.1] | 8.6 [5.3 to 12.9]
  Muscle pain: Moderate | 10.9 [7.2 to 15.6] | 9.9 [6.4 to 14.4]
  Muscle pain: Severe | 0.9 [0.1 to 3.1] | 0.9 [0.1 to 3.1]
  Joint pain: Any | 18.7 [13.9 to 24.3] | 18.0 [13.3 to 23.6]
  Joint pain: Mild | 9.1 [5.7 to 13.6] | 10.7 [7.1 to 15.4]
  Joint pain: Moderate | 9.1 [5.7 to 13.6] | 6.4 [3.6 to 10.4]
  Joint pain: Severe | 0.4 [0.0 to 2.4] | 0.9 [0.1 to 3.1]

79. Secondary Outcome: Stage1: Percentage of Participants With Antipyretic Medication Use 30 Days After Vaccination 1: Group 1 and Group 3
Time Frame: 30 days after Vaccination 1
Population: Vaccination 1 safety population included participants who received the first dose of investigational product (MenABCWY+saline or bivalent rLP2086+MenACWY-CRM) at Visit 1 (Month 0), and for whom safety information from Visit 1 (Month 0) to prior to Visit 3 (Month 6) was available. Here, 'Number of Participants Analyzed' signifies number of participants measured and analyzed for this outcome measure. Analysis was planned for Group 1 and Group 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 269 | 269
Percentage of participants | 20.8 [16.1 to 26.2] | 13.8 [9.9 to 18.5]

80. Secondary Outcome: Stage1: Percentage of Participants With Antipyretic Medication Use 30 Days After Vaccination 2: Group 1 and Group 3
Time Frame: 30 days after Vaccination 2
Population: Vaccination 2 safety population included participants who received the second dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 3 (Month 6), and for whom safety information from Visit 3 (Month 6) up to and including Visit 4 (month 7) was available. Here, 'Number of Participants Analyzed' signifies number of participants measured and analyzed for this outcome measure. Analysis was planned for Group 1 and Group 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 230 | 233
Percentage of participants | 17.8 [13.1 to 23.4] | 13.3 [9.2 to 18.4]

81. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 SAE Within 30 Days After Vaccination 1: Group 1 and Group 3
Description: as for outcome 9
Time Frame: 30 days after Vaccination 1
Population: Vaccination 1 safety population included participants who received the first dose of investigational product (MenABCWY+saline or bivalent rLP2086+MenACWY-CRM) at Visit 1 (Month 0), and for whom safety information from Visit 1 (Month 0) to prior to Visit 3 (Month 6) was available. Analysis was planned for Group 1 and Group 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 0.0 [0.0 to 1.3] | 0.7 [0.1 to 2.6]

82. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 SAE Within 30 Days After Vaccination 2: Group 1 and Group 3
Description: as for outcome 9
Time Frame: 30 days after Vaccination 2
Population: Vaccination 2 safety population included participants who received the second dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 3 (Month 6), and for whom safety information from Visit 3 (Month 6) up to and including Visit 4 (month 7) was available. Analysis was planned for Group 1 and Group 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 242 | 244
Percentage of participants | 0.4 [0.0 to 2.3] | 0.0 [0.0 to 1.5]

83. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 SAE Within 30 Days After Any Vaccination: Group 1 and Group 3
Description: as for outcome 9
Time Frame: 30 days after any vaccination
Population: The safety population for Stage 1 included participants who had received at least 1 dose of investigational product during Stage 1 and for whom safety data were available. Analysis was planned for Group 1 and Group 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 0.4 [0.0 to 2.0] | 0.7 [0.1 to 2.6]

84. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 SAE During the Vaccination Phase: Group 1 and Group 3
Description: as for outcome 9
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: Stage 1 safety population: participants who received at least 1 dose of investigational product during Stage 1 and for whom safety data were available. Analysis was planned for Group 1 and 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 0.4 [0.0 to 2.0] | 1.8 [0.6 to 4.3]

85. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 SAE During the Stage 1 Follow-up Phase: Group 1 and Group 3
Description: as for outcome 13
Time Frame: Stage 1 Follow-up phase: From 1 month after Vaccination 2 through 6 months after Vaccination 2 (5 Months)
Population: Stage 1 Follow-up Safety population: participants who received at least 1 dose of investigational product and for whom safety information was available from after Visit 4 (Month 7) up to and including Visit 5 (Month 12). Analysis was planned for Group 1 and 3 separately. Overall number of participants analysed included only those participants who met criteria for Stage 1 follow-up safety population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 239 | 239
Percentage of participants | 0.8 [0.1 to 3.0] | 0.4 [0.0 to 2.3]

86. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 SAE Throughout the Stage 1: Group 1 and Group 3
Description: as for outcome 13
Time Frame: Throughout Stage 1: From the Vaccination 1 through 6 months after Vaccination 2 (12 Months)
Population: Stage 1 safety population: participants who received at least 1 dose of investigational product during Stage 1 and for whom safety data were available. Analysis was planned for Group 1 and 3 separately. Here overall number of participants analysed included those participants who met criteria for Stage 1 safety population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 1.5 [0.4 to 3.7] | 2.2 [0.8 to 4.8]

87. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Vaccination 1: Group 1 and Group 3
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: 30 days after vaccination 1
Population: as for outcome 81
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 4.8 [2.6 to 8.0] | 5.9 [3.4 to 9.4]

88. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Vaccination 2: Group 1 and Group 3
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: 30 days after vaccination 2
Population: as for outcome 82
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 242 | 244
Percentage of participants | 5.8 [3.2 to 9.5] | 9.0 [5.7 to 13.3]

89. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Any Vaccination: Group 1 and Group 3
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: 30 days after any vaccination
Population: Stage 1 safety population: participants who received at least 1 dose of investigational product during Stage 1 and for whom safety data were available. Analysis was planned for Group 1 and Group 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 9.6 [6.3 to 13.7] | 13.3 [9.5 to 17.9]

90. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE During the Stage 1 Vaccination Phase: Group 1 and Group 3
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: as for outcome 84
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 23.9 [19.0 to 29.4] | 28.4 [23.1 to 34.2]

91. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE During the Stage 1 Follow-up Phase: Group 1 and Group 3
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Stage 1 Follow-up phase: From 1 month after Vaccination 2 through 6 months after Vaccination 2 (5 Months)
Population: Stage 1 Follow-up Safety population: participants who received at least 1 dose of investigational product and for whom safety information was available from after Visit 4 (Month 7) up to and including Visit 5 (Month 12). Analysis was planned for Group 1 and 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 239 | 239
Percentage of participants | 13.8 [9.7 to 18.8] | 18.8 [14.1 to 24.4]

92. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 Medically Attended AE Throughout the Stage 1: Group 1 and Group 3
Description: Medically attended AE was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Throughout Stage 1: From the Vaccination 1 through 6 months after Vaccination 2 (12 Months)
Population: as for outcome 84
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 30.9 [25.4 to 36.7] | 35.1 [29.4 to 41.1]

93. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 NDCMC Within 30 Days After Vaccination 1: Group 1 and Group 3
Description: as for outcome 21
Time Frame: 30 days after vaccination 1
Population: as for outcome 81
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 1.4]

94. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 NDCMC Within 30 Days After Vaccination 2: Group 1 and Group 3
Description: as for outcome 21
Time Frame: 30 days after vaccination 2
Population: as for outcome 82
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 242 | 244
Percentage of participants | 0.0 [0.0 to 1.5] | 0.0 [0.0 to 1.5]

95. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 NDCMC Within 30 Days After Any Vaccination: Group 1 and Group 3
Description: as for outcome 21
Time Frame: 30 days after any vaccination
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 1.4]

96. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 NDCMC During the Stage 1 Vaccination Phase: Group 1 and Group 3
Description: as for outcome 21
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 0.7 [0.1 to 2.6] | 0.0 [0.0 to 1.4]

97. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 NDCMC During the Stage 1 Follow-up Phase: Group 1 and Group 3
Description: as for outcome 21
Time Frame: Stage 1 Follow-up phase: From 1 month after Vaccination 2 through 6 months after Vaccination 2 (5 Months)
Population: Stage 1 Follow-up Safety population: participants who received at least 1 dose of investigational product and for whom safety information was available from after Visit 4 (Month 7) up to and including Visit 5 (Month 12). Analysis was planned for Group 1 and Group 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 239 | 239
Percentage of participants | 0.4 [0.0 to 2.3] | 0.0 [0.0 to 1.5]

98. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 NDCMC Throughout the Stage 1: Group 1 and Group 3
Description: as for outcome 21
Time Frame: Throughout Stage 1: From the Vaccination 1 through 6 months after Vaccination 2 (12 Months)
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 1.1 [0.2 to 3.2] | 0.0 [0.0 to 1.4]

99. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 AE Within 30 Days After Vaccination 1: Group 1 and Group 3
Description: as for outcome 27
Time Frame: 30 days after vaccination 1
Population: as for outcome 81
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 15.1 [11.0 to 19.9] | 11.1 [7.6 to 15.4]

100. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 AE Within 30 Days After Vaccination 2: Group 1 and Group 3
Description: as for outcome 27
Time Frame: 30 days after vaccination 2
Population: as for outcome 82
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 242 | 244
Percentage of participants | 16.1 [11.7 to 21.4] | 12.3 [8.5 to 17.1]

101. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 AE Within 30 Days After Vaccination Any Vaccination: Group 1 and Group 3
Description: as for outcome 27
Time Frame: 30 days after any vaccination
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 25.7 [20.6 to 31.4] | 19.9 [15.3 to 25.2]

102. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 AE During the Stage 1 Vaccination Phase: Group 1 and Group 3
Description: as for outcome 27
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 41.5 [35.6 to 47.6] | 36.9 [31.1 to 42.9]

103. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 Immediate AE After Vaccination 1: Group 1 and Group 3
Description: Immediate AE was defined as AE occurring within the first 30 minutes after investigational product administration.
Time Frame: 30 minutes after Vaccination 1
Population: Vaccination 1 safety population included participants who received the first dose of investigational product (MenABCWY+saline or bivalent rLP2086+MenACWY-CRM) at Visit 1 (Month 0), and for whom safety information from Visit 1 (Month 0) to prior to Visit 3 (Month 6) was available. Analysis was planned for Group 1 and 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Percentage of participants | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 1.4]

104. Secondary Outcome: Stage1: Percentage of Participants With at Least 1 Immediate AE After Vaccination 2: Group 1 and Group 3
Description: Immediate AE was defined as AE occurring within the first 30 minutes after investigational product administration.
Time Frame: 30 minutes after Vaccination 2
Population: Vaccination 2 safety population included participants who received the second dose of investigational product (MenABCWY or bivalent rLP2086) at Visit 3 (Month 6), and for whom safety information from Visit 3 (Month 6) up to and including Visit 4 (month 7) was available. Analysis was planned for Group 1 and 3 separately.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 242 | 244
Percentage of participants | 0.0 [0.0 to 1.5] | 0.0 [0.0 to 1.5]

105. Secondary Outcome: Stage1: Number of Participants Who Missed School/Work Due to AE During the Stage 1 Vaccination Phase: Group 1 and Group 3
Time Frame: Stage 1 Vaccination Phase: From Vaccination 1 through 1 month after Vaccination 2 (7 Months)
Population: Safety population for Stage 1 included participants who had received at least 1 dose of investigational product during Stage 1 and for whom safety data were available. Analysis was planned for Group 1 and Group 3 separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenABCWY + Saline (ACWY-Naive) | Group 3: MenABCWY + Saline (ACWY-Experienced)
Number analyzed (Participants) | 272 | 271
Participants | 38 | 46

ADVERSE EVENTS:
Time Frame: Systematic assessment: Local reactions and systemic events recorded within 7 days of each vaccination; Non-systematic collection: SAEs recorded from Month 0 to 6 months after Vaccination 2 (up to Month 12) and 6 months after Booster Vaccination (Booster Vaccination was at Month 54); Non-SAEs recorded from Month 0 to 1 month after Vaccination 2 ( up to Month 7); within 48 hours of blood draw at Month 18, 30 and 42; and 1 month after Booster Vaccination
Description: Same event may appear as both AE and SAE, but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety population for Stage 1: participants who received at least 1 dose of investigational product during Stage 1 and for whom safety data were available. Safety population for Stage 2: participants who received booster vaccination and for whom safety data were available.
Groups:
- Stage 1: Group 1: MenABCWY + Saline (ACWY-Naive); Stage 2: Group 1: MenABCWY + Saline (ACWY-Naive): Stage 1: ACWY-naive participants were randomized to receive an intramuscular injection of 0.5 milliliter (mL) of Neisseria meningitidis groups A, B, C, W, and Y vaccine (MenABCWY) and 0.5 mL of saline at Month 0, participants received 0.5 mL of MenABCWY vaccine intramuscularly at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received 0.5 mL of MenABCWY vaccine (booster vaccination) intramuscularly at Month 54.
- Stage 1: Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive); Stage 2: Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive): Stage 1: ACWY-naive participants were randomized to receive an intramuscular injection of 0.5 mL bivalent recombinant lipoprotein 2086 (rLP2086) vaccine and 0.5 mL of meningococcal group A, C, W-135, and Y conjugate vaccine (MenACWY-CRM) at Month 0. Participants received 0.5 mL of bivalent rLP2086 vaccine at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received intramuscularly injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL of MenACWY-CRM vaccine (booster vaccination) at Month 54.
- Stage 1: Group 3: MenABCWY + Saline (ACWY-Experienced); Stage 2: Group 3: MenABCWY + Saline (ACWY-Experienced): Stage 1: ACWY-experienced participants were randomized to receive an intramuscular injection of 0.5 milliliter (mL) of Neisseria meningitidis groups A, B, C, W, and Y vaccine (MenABCWY) and 0.5 mL of saline at Month 0, participants received 0.5 mL of MenABCWY vaccine intramuscularly at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received 0.5 mL of MenABCWY vaccine (booster vaccination) intramuscularly at Month 54.
- Stage 1: Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced); Stage 2: Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced): Stage 1: ACWY-experienced participants were randomized to receive an intramuscular injection of 0.5 mL bivalent recombinant lipoprotein 2086 (rLP2086) vaccine and 0.5 mL of meningococcal group A, C, W-135, and Y conjugate vaccine (MenACWY-CRM) at Month 0. Participants received 0.5 mL of bivalent rLP2086 vaccine at Month 6. Stage 1 was followed by Stage 2. Stage 2: Participants received intramuscularly injection of 0.5 mL of bivalent rLP2086 vaccine and 0.5 mL of MenACWY-CRM vaccine (booster vaccination) at Month 54.
Arm/Group | Stage 1: Group 1: MenABCWY + Saline (ACWY-Naive) | Stage 1: Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Stage 1: Group 3: MenABCWY + Saline (ACWY-Experienced) | Stage 1: Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced) | Stage 2: Group 1: MenABCWY + Saline (ACWY-Naive) | Stage 2: Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) | Stage 2: Group 3: MenABCWY + Saline (ACWY-Experienced) | Stage 2: Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced)
All-Cause Mortality (participants affected / at risk) | 1/272 | 0/534 | 0/271 | 0/523 | 0/114 | 0/65 | 0/101 | 0/73
Serious Adverse Events (participants affected / at risk) | 5/272 | 6/534 | 6/271 | 9/523 | 1/114 | 1/65 | 3/101 | 2/73
Other Adverse Events (participants affected / at risk) | 267/272 | 508/534 | 259/271 | 502/523 | 54/114 | 37/65 | 72/101 | 57/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Group 1: MenABCWY + Saline (ACWY-Naive) (N=272) | Stage 1: Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) (N=534) | Stage 1: Group 3: MenABCWY + Saline (ACWY-Experienced) (N=271) | Stage 1: Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced) (N=523) | Stage 2: Group 1: MenABCWY + Saline (ACWY-Naive) (N=114) | Stage 2: Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) (N=65) | Stage 2: Group 3: MenABCWY + Saline (ACWY-Experienced) (N=101) | Stage 2: Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced) (N=73)
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oppositional defiant disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Group 1: MenABCWY + Saline (ACWY-Naive) (N=272) | Stage 1: Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) (N=534) | Stage 1: Group 3: MenABCWY + Saline (ACWY-Experienced) (N=271) | Stage 1: Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced) (N=523) | Stage 2: Group 1: MenABCWY + Saline (ACWY-Naive) (N=114) | Stage 2: Group 2: Bivalent rLP2086 + MenACWY-CRM (ACWY-Naive) (N=65) | Stage 2: Group 3: MenABCWY + Saline (ACWY-Experienced) (N=101) | Stage 2: Group 4: Bivalent rLP2086 + MenACWY-CRM (ACWY-Experienced) (N=73)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pectus excavatum (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 1 | 2 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3 | 4 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 7 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 9 | 1 | 5 | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4 | 1 | 6 | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 4 | 11 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 3 | 3 | 2 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 6 | 5 | 2 | 13 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 6 | 2 | 13 | 2 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 4 | 4 | 2
Ear infection (Infections and infestations) | 3 | 6 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 6 | 14 | 4 | 9 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 8 | 12 | 4 | 6 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 9 | 14 | 4 | 18 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 11 | 19 | 16 | 21 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 3 | 2 | 2 | 5 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 11 | 6 | 4 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 3 | 5 | 1 | 2 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 9 | 8 | 15 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 6 | 9 | 9 | 13 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 5 | 9 | 9 | 14 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 2 | 7 | 6 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 32 | 11 | 28 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 11 | 5 | 10 | 1 | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 3 | 3 | 1 | 9 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 11 | 1 | 8 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 5 | 6 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 5 | 7 | 8 | 7 | 1 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 7 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 4 | 3 | 1 | 6 | 1 | 1 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 4 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 3 | 5 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 7 | 2 | 2 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 11 | 4 | 13 | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 5 | 3 | 1 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 7 | 3 | 2 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 6 | 0 | 5 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 4 | 4 | 1 | 4 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Psychophysiologic insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 6 | 0 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 4 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 3 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 0 | 4 | 4 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 3 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 6 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 55 | 104 | 54 | 105 | 3 | 4 | 7 | 7
Vomiting (Gastrointestinal disorders) | 13 | 31 | 13 | 33 | 2 | 0 | 2 | 1
Chills (General disorders) | 82 | 152 | 67 | 141 | 6 | 7 | 14 | 8
Fatigue (General disorders) | 180 | 315 | 163 | 344 | 28 | 24 | 47 | 37
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 256 | 479 | 251 | 480 | 48 | 34 | 65 | 50
Pyrexia (FEVER) (General disorders) | 29 | 56 | 17 | 37 | 3 | 1 | 0 | 1
Swelling (General disorders) | 77 | 123 | 67 | 114 | 11 | 9 | 14 | 10
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 79 | 153 | 78 | 148 | 12 | 10 | 16 | 9
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 104 | 204 | 87 | 186 | 11 | 12 | 24 | 13
Headache (Nervous system disorders) | 163 | 312 | 159 | 312 | 23 | 21 | 35 | 31
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 73 | 130 | 61 | 95 | 8 | 11 | 16 | 14

LIMITATIONS AND CAVEATS:
SAE of "pregnancy" for 1 participant during booster vaccination phase (Stage 2) was recorded erroneously and was reported in result of outcome measure 37.

One participant had an SAE which was recorded after 8 months of vaccination 2 and one participant had an SAE after 15 months of Vaccination 2. This time period did not present Stage 1 or Stage 2. Hence, it was not included in related outcome measure summary. However, these participants were included in adverse events module for Stage 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03135834/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT03135834/SAP_001.pdf